### STATISTICAL ANALYSIS PLAN

A Phase 1, Partially-Blinded, Placebo-Controlled, Randomized, Multiple Ascending Dose Study to Include A Single Dose Food-Effect Study to Evaluate the Safety, Tolerability, and the Pharmacokinetic Profile of TBI-223 in Healthy Adult Subjects

Global Alliance for TB Drug Development

Protocol No: TBI-223-CL-002

**TKL Study Number P1980121** 

TKL Research, Inc. One Promenade Blvd Fair Lawn, NJ 07410

24 March 2021

Jerry Nedelman, PhD
Senior Director, Pharmacometrics
Global Alliance for TB Drug Development

Michael Tuley, PhD Vice President, Data Sciences and Quality Assurance TKL Research, Inc.

| Jerry Redelman | | | | | | |
|---|---|---|---|---|---|---|
| Signer Name: Jerry Nedelman Signing Reason: I have reviewed this document Signing Time: April 20, 2021 8:04 AM PDT 7839E5A76523498AB928E27ED5F738EAPril | 20, | 2021 | 8 | 8:04 | АМ | P |
| Signature | D | ate | | | | |
| DocuSigned by: Midual Tidey Signer Name: Michael Tuley Signing Reason: I approve this document Signing Time: April 20, 2021 8.07 AM PDT BE981D7A319443499E30D520D1EBB3F | 1 20 | , 2021 | 1 | 8:07 | ' AM | 1 |
| Signature | D | ate | | _ | | |

### **Table of Contents**

| Tab | e of Contents | 2 |
|------|----------------------------------------------------|----|
| List | of Abbreviations and Definitions of Terms | .4 |
| 1. | NTRODUCTION | 6 |
| 2. | STUDY OBJECTIVES | 6 |
| 3. | STUDY DESIGN | |
| 4. | HARDWARE AND SOFTWARE | |
| 5. | STATISTICAL DATA REVIEW | .8 |
| 6. | DATABASE CLOSURE | 8 |
| 7. | SAMPLE SIZE DETERMINATION | 8 |
| 8. | HANDLING OF MISSING DATA | 8 |
| 9. | ANALYSIS POPULATIONS | |
| | 3.1 Safety Population | |
| | 3.2 Pharmacokinetic (PK) Population | |
| 10. | DATA CONVENTIONS FOR ANALYSIS | |
| | 0.1 General Statistical Principles | 9 |
| | 0.2 Study Day | |
| 11. | STATISTICAL EVALUATION | 10 |
| | 0.1 Subject Disposition | 10 |
| | 0.2 Demographic and Other Baseline Characteristics | 10 |
| | 0.3 Study Drug Administration | 10 |
| | 0.4 Prior and Concomitant Medications | 10 |
| | 0.5 Medical History | 11 |
| | 0.6 Efficacy Analysis | 11 |
| | 0.7 Safety Analysis | 11 |
| | 0.7.1 Adverse and Serious Adverse Events | 11 |
| | 0.7.2Clinical Laboratory Tests | 12 |

| | 10.7.3 Electrocardiogram | 12 |
|-----|-------------------------------------------------|----|
| | 10.7.4Vital Signs | 12 |
| | 10.7.5 Physical Examination. | 13 |
| | 10.8 Pharmacokinetic Analysis | 13 |
| 12. | CHANGES FROM THE PROTOCOL AND PLANNED ANALYSES | 15 |
| 13. | HEADINGS | 15 |
| 14. | ARCHIVING AND RETENTION OF DOCUMENTS | 16 |
| 15. | REFERENCES | 16 |
| 16 | OUTLINE OF PROPOSED TABLES FIGURES AND LISTINGS | 16 |

### **List of Abbreviations and Definitions of Terms**

| Abbreviation | Definition |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AI | Accumulation Index |
| ANOVA | Analysis of Variance |
| AUC | Area under the plasma concentration versus time curve |
| $\mathrm{AUC}_{\mathrm{inf}}$ $\mathrm{AUC}_{0\text{-}24}$ | Area under the plasma concentration versus time curve from Time 0 to infinity (by extrapolation); also reported as AUC <sub>(0-inf)</sub> Area under the plasma concentration versus time curve from Time 0 to |
| BMI | the end of the dosing period Body Mass Index |
| BP | Blood Pressure |
| BPM | Beats Per Minute |
| C | Celsius (Centigrade) |
| CI | Confidence Interval |
| CL/F | Apparent Oral Clearance |
| $C_{max}$ $C_{min}$ | Observed Maximum Plasma Concentration Observed Minimum Plasma Concentration |
| CS | Clinically Significant |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| DBP | Diastolic Blood Pressure |
| DIC | Drug-in-Capsule |
| DMP | Data Management Plan |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| FDA | US Food and Drug Administration |
| GMR | Geometric Mean Ratio |
| IL-17 | Interleukin-17 |
| $\lambda_{\mathrm{z}}$ | Elimination Rate Constant |
| kg | Kilogram |
| mg | Milligram |

| Abbreviation | Definition |
|---|---|
| mL | Milliliter |
| msec | Millisecond |
| ODS | Output Delivery System |
| N/A | Not Applicable |
| NCS | Not Clinically Significant |
| PD | Pharmacodynamics |
| PK | Pharmacokinetics |
| PR | Duration between the beginning of the P wave and the beginning of the next QRS complex on the ECG |
| PT | Preferred Term |
| QRS | Duration between the start of the Q wave and the end of the S wave on the ECG. Also known as ventricular depolarization complex. |
| QT | Duration between the start of the Q wave and the end of the T wave on the ECG |
| QTc | QT interval corrected for heart rate |
| QTcB | Corrected QT interval using Bazett's Formula |
| QTcF | Corrected QT interval using Fridericia's Formula |
| RTF | Rich-Text Format |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SBP | Systolic Blood Pressure |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| TEAE | Treatment-Emergent Adverse Event |
| $t_{1/2}$ | Half-life |
| $T_{\text{max}}$ | Time at which C <sub>max</sub> occurs |
| $T_{\min}$ | Time at which C <sub>min</sub> occurs |
| V <sub>z</sub> /F | Apparent Volume of Distribution |

### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the study Protocol Version 1.0 dated 04 December 2020. This document specifies, prior to locking the database, a comprehensive description of the rationale, strategies, and statistical techniques that are planned to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of multiple dose TBI-223 in normal healthy volunteers.

This document also provides additional details concerning the statistical analyses outlined in the protocol and reflects any changes to the protocol from any amendments. This plan will not repeat all the definitions given in the protocol but will provide further details of the summaries and analyses planned therein.

### 2. STUDY OBJECTIVES

The primary objective of the study is to evaluate the safety and tolerability of multiple doses of TBI-223 in healthy adult subjects.

The secondary objective of the study is:

- To determine the pharmacokinetics (PK) of TBI-223 and its metabolite, M2 after multiple ascending doses of TBI-223 in healthy adult subjects when administered after a high-calorie, high-fat meal
- For the TBI-223 sustained-release (SR1) formulation and for the combination of the SR and immediate-release (IR) formulations, to compare the PK profiles of a single dose when administered to healthy adult subjects in the fasting state versus after a high-calorie, high-fat meal
- To determine the pharmacokinetics (PK) of a single dose of the TBI-223 sustained-release (SR1) formulation in healthy adult subjects when administered fasted

### 3. STUDY DESIGN

This is a partially-blinded, placebo-controlled, randomized multiple ascending dose (MAD) study to be conducted at one study center.

Thirty-six (36) subjects will be enrolled in 3 cohorts with 12 subjects per cohort. Within each cohort, 9 subjects will be assigned to receive active treatment and 3 subjects will receive placebo. Each subject will participate in one dose level.

The first 2 cohorts (food-effect cohorts) will begin dosing of TBI-223 on Day 1 under fasted conditions, followed by a 3 day washout period and then by multiple doses of TBI-223

administered after a high-calorie, high-fat meal from Day 4 through Day 17 (total of 14 days). The third cohort (non-food-effect cohort) will begin dosing of TBI-223 on Day 1 and continue through Day 14, all doses administered after a high-calorie, high-fat meal.

Each subject will be administered TBI-223 tablets (SR1 or IR or a combination of both formulations) or placebo once daily for 14 days with corresponding pharmacokinetic measurements. After each dose cohort, the Sponsor and Investigator will review the pharmacokinetic and safety data before proceeding to the next dose level.

Dose escalation to the next cohort (i.e., dose level) or decisions regarding changed or additional cohorts will not take place until the Sponsor, in conjunction with the Principal Investigator and dose escalating committee, has determined that adequate safety, tolerability, and pharmacokinetics from the previous cohort(s) have been demonstrated to permit proceeding to the next cohort. The Institutional Review Board (IRB) should be immediately notified of the dose escalation or any revised approach for review and approval.

Safety will be assessed throughout the study for all subjects. Safety assessments will include physical and detailed neurological examinations, vital signs (blood pressure, pulse rate, respiration rate, temperature and pulse oximetry), electrocardiograms (ECGs), cardiac monitoring, adverse events (AEs), and clinical laboratory tests (including hematology, serology, serum chemistry, coagulation, and urinalysis).

Blood and urine will be collected for clinical laboratory evaluations.

The Principal Investigator, in conjunction with the Sponsor may collect additional blood if necessary, for repeat laboratory or safety evaluations including AE follow up.

Female subjects will have blood collected for serum pregnancy testing. Females claiming postmenopausal status will have blood collected to measure follicle stimulating hormone (FSH) levels.

During each cohort, blood samples (trough samples) will be obtained before each dose of study drug, and at the time points on the events schedule. Plasma pharmacokinetic samples will be analyzed for TBI-223 and M2 using validated analytical methods. Appropriate pharmacokinetic parameters will be calculated using non compartmental methods.

### 4. HARDWARE AND SOFTWARE

Statistical analysis will be performed following TKL standard operating procedures and on the TKL computer network. All statistical analyses will be performed using SAS Version 9.4 or higher with program code prepared specifically for the project by qualified TKL statisticians and SAS programmers.

The SAS programs will generate rich-text-formatted (RTF) output with the "RTF" extension using the SAS Output Delivery System (ODS). The summary tables and listings will be formatted using the Times New Roman font. The RTF output is included in report documents prepared with Microsoft Word and converted to PDF format without typographical change.

Study data tabulation model (SDTM) data sets and required analysis data model (ADaM) data sets will be created and taken as input to validated SAS programs to generate the report-ready tables, listings, and figures. Each output display will show the names of the data sets and SAS program used to produce it. Upon completion of the study report, the data sets will be provided to the sponsor as SAS XPT transport files with define.xml files including details of all derivations and imputations used.

### 5. STATISTICAL DATA REVIEW

Data verification activities to be performed prior to delivery of the SAS data sets to the project statistician are described in the approved Data Management Plan (DMP). After completion of the data verification activities, the SAS data sets will be reviewed by the project statistician along with documentation of any unresolved queries and data conventions applied that are not fully explained in the data or in the DMP. The project statistician will perform completeness and self-consistency checks of the study data. Questions will be issued to the Data Manager and resolved before closure of the database.

### 6. DATABASE CLOSURE

After completion of all data review procedures, validation of the project database, and approval of the data review document by the study sponsor, the clinical database will be closed, termed "Database Lock". Any change to the clinical database after this time will require written authorization, with explanation, by the Sponsor and the Biostatistician.

### 7. SAMPLE SIZE DETERMINATION

The sample size and the number of subjects for each cohort is expected to provide sufficient safety and tolerability data to evaluate whether escalation to the next dose level is warranted. This study has not been formally powered and the sample size was not based on statistical considerations.

### 8. HANDLING OF MISSING DATA

No imputation is planned for safety data unless otherwise specified below. All efforts will be made to ensure completeness for AE severity and AE drug-relationship data.

The handling of any missing drug concentration-time data to estimate PK parameters is described in the PK analysis section.

### 9. ANALYSIS POPULATIONS

Two populations will be defined for analysis detailed in this document: the Safety Population and the PK Population.

### 8.1 Safety Population

The Safety Population will include all randomized subjects who receive at least one dose of the study drugs (TBI-223 or placebo). Subjects will be analyzed according to the treatment subjects actually received regardless of the treatment to which they were randomized. Subjects who receive placebo will be pooled across dosing panels to form a single placebo group.

### 8.2 Pharmacokinetic (PK) Population

All subjects who receive TBI-223 and who have plasma concentration data available will be included in the PK population. This population will be used for the presentation of plasma concentration results as well as PK analysis. However, only subjects with profiles adequate to determine PK parameters will be included in PK analyses, which will be decided by a PK scientist upon review of all concentration profiles.

### 10. DATA CONVENTIONS FOR ANALYSIS

### 9.1 General Statistical Principles

All statistical processing will be performed using the SAS system (Version 9.4 or higher). The focus of the statistical analysis will be to assess the safety, tolerability, and PK of TBI-223 in normal healthy volunteers.

Descriptive statistics will be used to provide an overview of the safety and PK results. For categorical parameters, the number and percentage of subjects in each category will be presented. The denominator for percentage will be based on the number of subjects appropriate for the purpose of analysis. For continuous parameters, descriptive statistics will include n (number of subjects), mean, standard deviation (SD), median, and range. In addition, coefficient of variation (%CV) and geometric mean will also be reported for appropriate PK parameters.

### 9.2 Study Day

Day 1 is defined as the date of first study drug administration. The day before Day 1 is Day -1; there is no Day 0. Study day is calculated relative to the date of Day 1.

Baseline is defined as the last available measurement prior to the first dose of the study drug on Day 1.

### 11. STATISTICAL EVALUATION

### 10.1 Subject Disposition

A subject disposition table will present the number of subjects screened, randomized, completed, and discontinued, along with the primary reason for discontinuation, as well as the number of subjects within each population. The summary will be presented for each TBI-223 dose, an "Any TBI-223" group including subjects receiving any TBI-223, and a pooled placebo group.

A listing of the subjects who are enrolled, randomized, and who complete or discontinue the study, along with the reason for and day of discontinuation, will be provided. Screen failures and protocol deviations will be presented in by-subject listings.

### 10.2 Demographic and Other Baseline Characteristics

The following demographic and baseline variables will be listed and summarized by treatment(TBI-223 by dose, any TBI-223, and pooled placebo) and overall:

- Age (years)
- Sex
- Race (American Indian or Alaskan Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, White, Multiple)
- Ethnicity origin (Hispanic or Latino, Not Hispanic or Latino)
- Weight (kg)
- Height (cm)
- BMI (kg/m<sup>2</sup>)

For continuous variables, descriptive statistics (mean, standard deviation, median, minimum, and maximum) will be provided. For categorical variables, the number and frequency of subjects in each category (sex, ethnicity, race) will be provided.

### 10.3 Study Drug Administration

A summary table for drug exposure will be provided by treatment (TBI-223 by dose, any TBI-223, and pooled placebo), and will include the number and percentage of subjects who receive at least one dose, at least one dose under fed conditions, all intended (i.e., 14 or 15) doses, as well as each single-dose treatment on each day. In addition, descriptive statistics (mean, standard deviation, median, minimum, and maximum) will be provided for the total number of doses for each dose group. A by-treatment, by-subject listing will be provided for date and time of each dose of study drug.

### 10.4 Prior and Concomitant Medications

Records of prior (with stop dates prior to Day 1) and concomitant medications (with stop dates on or after Day 1) will be provided in a by-treatment, by-subject listing.

### 10.5 Medical History

Current conditions and past medical conditions will be provided in a by-treatment, by-subject listing.

### 10.6 Efficacy Analysis

No efficacy analysis or hypothesis testing will be performed.

### 10.7 Safety Analysis

All safety analyses are based on the Safety Population according to the actual study drug and dose received. Detailed analyses will be described in sections below.

The following safety endpoints will be summarized:

- Adverse Events;
- Clinical safety laboratory testing;
- Standard 12-lead ECG data;
- Physical examinations;
- Vital signs

Interim analyses of safety results from each panel before dose escalation will be reviewed by the Investigator and Medical Monitor, but will not be analyzed statistically.

### 10.7.1 Adverse and Serious Adverse Events

AE terms will be coded using the MedDRA version 23.1 (2020) dictionary. A treatment-emergent AE (TEAE) is defined as an AE with a start date and time coinciding with or after the first dose of study drug received.

All AEs will be presented in a by-treatment, by-subject, detailing the verbatim term given by the investigator, the preferred term (PT), system organ class (SOC), onset date and time, end date and time, severity, outcome, relationship to study drug, action taken with study drug, other action taken, seriousness and criteria for seriousness. Serious AEs and AEs leading to study discontinuation will also be presented in a separate listing.

An overall summary of TEAEs will be presented by treatment (TBI-223 by dose, any TBI-223, and pooled placebo). The summary will include the total number of events, frequency counts and percentages with:

- Any TEAE
- Any serious TEAE
- Any treatment-related TEAE (that is, TEAEs that are probably and possibly related)
- Any treatment-related serious TEAE
- Any TEAE resulting in withdrawal from the study
- Any deaths

Summaries of the incidence of the following TEAEs will be displayed by treatment (TBI-223 by dose, any TBI-223, and pooled placebo):

- All TEAEs by PT in descending order of frequency of any TBI-223
- All treatment-related TEAEs by PT in descending order of frequency of any TBI-223
- All TEAEs by SOC, PT, and maximum severity (mild, moderate, or severe)
- All treatment-related TEAEs by SOC, PT, and maximum severity
- All TEAEs by SOC, PT, and maximum causality (not related, possible, probably) to the study drug

For purpose of the summary of the incidence, each subject will contribute only once (i.e., the first occurrence, the occurrence with the maximum severity or causality) within an SOC and a PT, regardless of the number of occurrences (events) the subjects experiences.

### 10.7.2 Clinical Laboratory Tests

Data listings by-treatment and by-subject will be provided for all laboratory parameters. Absolute values and changes from baseline will also be summarized for hematology and clinical chemistry parameters using descriptive statistics by treatment at the following time points: Baseline, Days 3, 5, 9, 10, 11 and follow-up visit).

Normal ranges and values outside the normal ranges will be identified by the central laboratory. A separate listing of out of normal range laboratory results will be provided. Shift tables will be provided for the number of subjects with clinical laboratory values below, within, or above normal ranges at each post-baseline visit relative to baseline, for each test.

Serum pregnancy, drug, alcohol, and cotinine screening results will be presented in a by-treatment, by-visit, by-subject listing.

### 10.7.3 Electrocardiogram

Tabulation of standard 12-lead ECG numeric results (ventricular rate, PR, QRS, QT, QTcF intervals) will be presented using descriptive statistics by treatment (TBI-223 by dose, any TBI-223, and pooled-placebo) for absolute values and changes from baseline for the following time points: Baseline, Day 1 post-dose, Day 4 post-dose, Day 14 or 17 pre-dose and post dose, and final assessment.

The number and percentage of subjects with post-baseline values of >450, >480, and >500 msec, as well as subjects with change from baseline of >30 (including subjects with >60 msec changes) and >60 msec at any post-baseline time point will be summarized for QTcF intervals.

Any clinically significant ECG results were to be captured as AEs by the PI. A by-treatment and by-subject listing of standard ECG results (numeric results and verbatim findings) will also be presented.

### 10.7.4 Vital Signs

Vital signs data will be presented in a by-treatment and by-subject listing for the following tests:

- Blood pressure (mmHg) both systolic and diastolic
- Pulse rate (beats per min)
- Respiration rate (breaths per min)
- Body temperature (°C)
- Pulse Oximetry

Absolute values and changes from baseline (i.e., the last available measurement prior to Day 1 dosing) will be summarized using descriptive statistics by treatment for the following time points:

- Baseline
- Day 1 6 hours post-dose
- Days 4 17 or 2 to 14 pre-dose
- Day 17 or 14 pre-dose
- Day 17 or 14 6 hours post-dose, change from Day 4 or Day 2 pre-dose value will also be summarized
- Follow-up visits

### 10.7.5 Physical Examination

Physical examination results will be presented in a by-subject listing. Clinically significant physical examination results will be reported as AEs by the PI.

### 10.8 Pharmacokinetic Analysis

All analyses of pharmacokinetics (PK) will be based on the PK population. Plasma concentrations of TBI-223 and M2 will be listed and summarized by cohort for each nominal time point, giving number of subjects, mean, standard deviation, median, minimum, maximum, and coefficient of variation [CV]). Mean and individual concentrations (TBI-223 and M2) will be plotted versus time for each cohort, for the following time periods:

- 0 to 24 h post-dose, Cohorts 1 and 2, Days 1, 4, and 17, linear and semi-log scales
- 0 to 24 h post-dose, Cohort 3, Days 1 and 14, linear and semi-log scales
- 0 to 72 h post-dose, Cohorts 1 and 2, Days 1 and 17, linear and semi-log scales
- 0 to 72 h post-dose, Cohort 3, Day 14, linear and semi-log scales
- Trough (Pre-dose and 24 h) Concentrations (Approach to Steady State), Cohorts 1 and 2, Days 4 to 17
- Trough (Pre-dose and 24 h) Concentrations (Approach to Steady State), Cohort 3, Days 1 to 14

Pharmacokinetic parameters for TBI-223 and M2 will be calculated as defined in Table 1 below. Only subjects with measured concentrations adequate to determine PK parameters will be included in the PK analyses.

**Table 1: Pharmacokinetic Parameters** 

| PK<br>parameter | Definition | Scope |
|---|---|---|
| C <sub>max</sub> | Maximum plasma concentration | [a] |
| AUC <sub>0-24</sub> | Area under the concentration curve from 0 to 24 h post-dose, calculated by trapezoidal integration | [a] |
| AUCinf | Area under the concentration curve extrapolated to complete elimination, calculated as $AUC_{inf} = AUC_{last} + \frac{c_{last}}{\lambda_z}$ where | [b] |
| | C <sub>last</sub> is the last measured post-dose concentration. | |
| $T_{\text{max}}$ | Time of the maximum plasma concentration, given as the nominal time point | [a] |
| C <sub>min</sub> | Minimum concentration during dosing period at steady state | [d] |
| T <sub>min</sub> | Time of minimum concentration during dosing period at steady state | [d] |
| C <sub>trough</sub> | Trough concentrations (pre-dose or 24-hour) | [c] |
| $\lambda_{\rm z}$ | Elimination rate constant, calculated as the slope of log-<br>transformed concentration vs time during the elimination<br>phase. | [a] |
| t <sub>1/2</sub> | Elimination half-life, calculated as $\frac{\ln 2}{\lambda_z}$ | [a] |
| CL/F | Apparent plasma drug clearance, calculated as $\frac{Dose}{AUC_{0-inf}}$ | [b] |
| CL <sub>ss</sub> /F | Apparent plasma drug clearance at expected steady state, calculated as $\frac{Dose}{AUC_{0-24}}$ | [d] |
| V <sub>Z</sub> /F | Apparent volume of distribution, calculated as $\frac{CL/F}{\lambda_z}$ | [b] |
| V <sub>zss</sub> /F | Apparent volume of distribution at expected steady state, calculated as $\frac{CL_{ss}/F}{\lambda_z}$ | [d] |
| R <sub>AUC</sub> , R <sub>Cmax</sub> | Accumulation ratio for $AUC_{0-24}$ ( $C_{max}$ ) calculated as the ratio of the value at steady state to the value during the first dosing period. | |

<sup>[</sup>a] Days 1, 4, and 17 (Cohorts 1 and 2); Days 1 and 14 (Cohort 3)

<sup>[</sup>b] Days 1 and 4 (Cohorts 1 and 2); Day 1 (Cohort 3)

<sup>[</sup>c] All dosing days

<sup>[</sup>d] Day 17 (Cohorts 1 and 2); Day 14 (Cohort 3)

Actual sample collection times will be used for the purpose of calculating PK parameters. Concentration data below the limit of quantitation (BLQ) will be marked as such in the data listings; they will be imputed as 0 for the calculations of descriptive statistics and for calculation of AUC<sub>0-24</sub>. Parameters will be presented in by-subject listings and summarized by dose group using mean, standard deviation, median, minimum, and maximum, as well as coefficient of variation and geometric mean for appropriate parameters.

The elimination rate constant will be estimated by linear regression using no fewer than 3 sampling points during the elimination phase. The first sampling time to be included in the calculation will be determined by visual inspection of the by-subject plots.

The food effect will be estimated for  $AUC_{0-24}$ ,  $AUC_{inf}$ , and  $C_{max}$  in Cohorts 1 and 2 by the ratio of geometric means of Day 4 (fed) to Day 1 (fasted) values. These will be presented along with the 90% 2-sided confidence intervals. These estimates will be calculated for each dose level using analysis of variance of the log-transformed values including the effects of subject and day. The differences of the least-squares means and confidence limits will then be back-transformed to provide the ratios of geometric means and their confidence limits. The food effect on  $T_{max}$  will be compared using the Wilcoxon Signed Rank test.

The achievement of steady state will be confirmed through analysis of trough (pre-dose / 24-hour concentrations) from Days 7 through 14 (Cohort 3) or Days 10 through 17 (Cohorts 1 and 2). (The 24-hour concentration for Day 17 may be used as a trough concentration at the end of the last dosing period.) These values will be analyzed in each cohort using analysis of variance with effects of subject and day (taking day as a 1-degree-of-freedom regressor effect, ie, not in the CLASS statement). If the effects of day and subject-day interaction are not found to be significant at the 5% level, then steady state will have been achieved. (Note that failure to reject the null hypothesis of the 5% 2-sided test of the effect of day in the proposed regression model is equivalent to a finding that the 95% 2-sided confidence limit on the slope includes the value 0.)

In a supplemental exploratory analysis, the values of  $AUC_{0-24}$  and  $C_{max}$  will be analyzed for differences between males and females. This analysis will be performed separately for each cohort and study day (8 separate analyses for each parameter) using by-gender summary statistics and 2-sample t tests.

### 12. CHANGES FROM THE PROTOCOL AND PLANNED ANALYSES

There are no major changes to the planned analyses as stated in the protocol. Any minor changes were for the purpose of streamlining the analysis.

### 13. HEADINGS

Each page of the analysis will show the sponsor's name, the investigational product, and the protocol number. Report tables will be embedded in the MS Word report document from SAS program output without change. The footer of each table will show the name of the SAS program

module which generated it, the names of all data sets providing input data in the program and the date and time the table was generated.

### 14. ARCHIVING AND RETENTION OF DOCUMENTS

After finalization of the analysis, the following will be archived at TKL Research, Inc. and/or with the study sponsor:

- SAP and any amendments
- DMP and Database Specification
- All SAS code used in the project for statistical analysis, report tables generation, and analysis data set creation
- Tables, listings and figures as included in the clinical study report
- SAS study data tabulation model (SDTM) and analysis dataset model (ADaM) datasets
- Relevant correspondence
- Any other pertinent study document (i.e. study protocol, investigator's brochure, correspondence, study report(s), etc.).

### 15. REFERENCES

No references are included.

### 16. OUTLINE OF PROPOSED TABLES, FIGURES AND LISTINGS

All the mock-up shells will be included in a separate document.

## 15. OUTLINE OF PROPOSED TABLES, FIGURES AND LISTINGS

### **Summary Tables**

| 14.1 | Summary of Disnosition Demographic and Evnosure Tables |
|---|---|
| | cummant of Disposition, Demographic, and Daposition Tables |
| | Summary of Subject Disposition |
| 14.1.2 | Summary of Subject Demographics and Baseline Characteristics |
| 14.1.3.1 | Summary of Extent of Exposure to TBI-223 |
| 14.2 | Summary of Pharmacokinetics Tables |
| 14.2.1.1 | Summary of Plasma TBI-223 and M2 Concentration (ng/mL) by Time Point, TBI-223 1800mg |
| 14.2.1.2 | Summary of Plasma TBI-223 and M2 Concentration (ng/mL) by Time Point, TBI-223 2400mg |
| 14.2.1.3 | Summary of Plasma TBI-223 and M2 Concentration (ng/mL) by Time Point, TBI-223 3000mg |
| 14.2.2.1.1 | Summary of TBI-223 Pharmacokinetic Parameters, Day 1 and Day 17, TBI-223 1800mg |
| 14.2.2.1.2 | Summary of TBI-223 Pharmacokinetic Parameters, Day 1 and Day 17, TBI-223 2400mg |
| 14.2.2.2.1 | Summary of TBI-223 Pharmacokinetic Parameters, Day 4 and Day 17, TBI-223 1800mg |
| 14.2.2.2.2 | Summary of TBI-223 Pharmacokinetic Parameters, Day 4 and Day 17, TBI-223 2400mg |
| 14.2.2.2.3 | Summary of TBI-223 Pharmacokinetic Parameters, Day 1 and Day 14, TBI-223 3000mg |
| 14.2.3 | Summary of TBI-223 Pharmacokinetic Parameters, Food Effect |
| 14.2.4 | Summary of TBI-223 Pharmacokinetic Parameters, Confirmation of Steady State |
| 14.2.5 | Summary of TBI-223 Pharmacokinetic Parameters, Analysis of Gender Differences |
| 14.2.6.1.1 | Summary of M2 Pharmacokinetic Parameters, Day 1 and Day 17, TBI-223 1800mg |
| 14.2.6.1.2 | Summary of M2 Pharmacokinetic Parameters, Day 1 and Day 17, TBI-223 2400mg |
| 14.2.6.2.1 | Summary of M2 Pharmacokinetic Parameters, Day 4 and Day 17, TBI-223 1800mg |
| 14.2.6.2.2 | Summary of M2 Pharmacokinetic Parameters, Day 4 and Day 17, TBI-223 2400mg |
| 14.2.6.2.3 | Summary of M2 Pharmacokinetic Parameters, Day 1 and Day 14, TBI-223 3000mg |
| 14.2.7 | Summary of M2 Pharmacokinetic Parameters, Food Effect |
| 14.2.8 | Summary of M2 Pharmacokinetic Parameters, Confirmation of Steady State |
| 14.2.9 | Summary of M2 Pharmacokinetic Parameters, Analysis of Gender Differences |

| 14.3 | Summary of Safety Tables |
|---|---|
| 14.3.1.1 | Overall Summary of Treatment-Emergent Adverse Events by Treatment |
| 14.3.1.2 | Summary of Treatment-Emergent Adverse Events by Preferred Term in Descending Frequency |
| 14.3.1.3 | Summary of Treatment-Related Treatment-Emergent Adverse Events by Preferred Term in Descending Frequency |
| 14.3.1.4 | Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term by Maximum Severity |
| 14.3.1.5 | Summary of Treatment-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term by Maximum Severity |
| 14.3.1.6 | Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term by Maximum Causality |
| 14.3.2.1.1 | Summary of Clinical Hematology: Absolute Values and Change from Baseline by Treatment and Time Point; Safety Population |
| 14.3.2.1.2 | Summary of Clinical Chemistry: Absolute Values and Change from Baseline by Treatment and Time Point; Safety Population |
| 14.3.2.1.3 | Summary of Clinical Coagulation: Absolute Values and Change from Baseline by Treatment and Time Point; Safety Population |
| 14.3.2.2.1 | Summary of Clinical Hematology: Categorical Change from Baseline |
| 14.3.2.2.2 | Summary of Clinical Chemistry: Categorical Change from Baseline |
| 14.3.2.2.3 | Summary of Clinical Coagulation: Categorical Change from Baseline |
| 14.3.2.3.1 | Summary of Laboratory Values Outside of Normal Range and Investigator's Assessment; Hematology |
| 14.3.2.3.2 | Summary of Laboratory Values Outside of Normal Range and Investigator's Assessment; Chemistry |
| 14.3.2.3.3 | Summary of Laboratory Values Outside of Normal Range and Investigator's Assessment; Coagulation |
| 14.3.2.4.1 | Summary of 12-Lead ECG Numeric Results; Absolute Values and Change from Baseline by Treatment and Visit; Safety Population |
| 14.3.2.4.2 | Summary of 12-Lead ECG Categorical Analysis, QTcF, Safety Population |
| 14.3.2.5 | Summary of Vital Signs; Absolute Values and Change from Baseline by Treatment and Time point; Safety Population |

### Figures

### 14.2.A.1.11-14.2.A.1.3.2

Mean TBI-223 Plasma Concentration by Treatment and Time Point, 0 to 24 Hours Post-dose

| 14.2.A.1.1.1 | Mean TBI-223 Plasma Concentration by Treatment and Time Point, Linear Scale<br>Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state)<br>Cohort 1, PK Population |
|---|---|
| 14.2.A.1.1.2 | Mean TBI-223 Plasma Concentration by Treatment and Time Point, Log-linear Scale<br>Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state)<br>Cohort 1, PK Population |
| 14.2.A.1.2.1 | Mean TBI-223 Plasma Concentration by Treatment and Time Point, Linear Scale<br>Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state)<br>Cohort 2, PK Population |
| 14.2.A.1.2.2 | Mean TBI-223 Plasma Concentration by Treatment and Time Point, Log-linear Scale Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state) Cohort 2, PK Population |
| 14.2.A.1.3.1 | Mean TBI-223 Plasma Concentration by Treatment and Time Point, Linear Scale<br>Hours 0 to 24 Post-Dose, Days 1 (single dose) and 14 (steady state)<br>Cohort 3, PK Population |
| 14.2.A.1.3.2 | Mean TBI-223 Plasma Concentration by Treatment and Time Point, Log-linear Scale<br>Hours 0 to 24 Post-Dose, Days 1 (single dose) and 14 (steady state)<br>Cohort 3, PK Population |

### 14.2.A.2.1.1-14.2.A.2.3.2

Mean TBI-223 Plasma Concentration by Treatment and Time Point, 0 to 72 Hours Post-dose

| 14.2.A.2.1.1 | Mean TBI-223 Plasma Concentration by Treatment and Time Point, Linear Scale<br>Hours 0 to 72 Post-Dose, Days 1 (single dose, fasted) and 17 (steady state, fed)<br>Cohort 1, PK Population |
|---|---|
| 14.2.A.2.1.2 | Mean TBI-223 Plasma Concentration by Treatment and Time Point, Log-linear Scale<br>Hours 0 to 72 Post-Dose, Days 1 (single dose, fasted) and 17 (steady state, fed)<br>Cohort 1, PK Population |

| 14.2.A.2.2.1 | Mean TBI-223 Plasma Concentration by Treatment and Time Point, Linear Scale Hours 0 to 72 Post-Dose, Days 1 (single dose, fasted) and 17 (steady state, fed) Cohort 2, PK Population |
|---|---|
| 14.2.A.2.2.2 | Mean TBI-223 Plasma Concentration by Treatment and Time Point, Log-linear Scale<br>Hours 0 to 72 Post-Dose, Days 1 (single dose, fasted) and 17 (steady state, fed)<br>Cohort 2, PK Population |
| 14.2.A.2.3.1 | Mean TBI-223 Plasma Concentration by Treatment and Time Point, Linear Scale<br>Hours 0 to 72 Post-Dose, Day 14 (steady state)<br>Cohort 3, PK Population |
| 14.2.A.2.3.2 | Mean TBI-223 Plasma Concentration by Treatment and Time Point, Log-linear Scale<br>Hours 0 to 72 Post-Dose, Day 14 (steady state)<br>Cohort 3, PK Population |

### 14.2.A.3.1-14.2.A.3.3

## Mean TBI-223 Plasma Trough Concentration by Treatment and Time Point, Approach to Steady State

| 14.2.A.3.1 | Mean TBI-223 Plasma Trough Concentrations by Treatment and Time Point, Approach to Steady State, Days 4 to 17<br>Cohort 1, PK Population |
|---|---|
| 14.2.A.3.2 | Mean TBI-223 Plasma Trough Concentrations by Treatment and Time Point, Approach to Steady State, Days 4 to 17 Cohort 2, PK Population |
| 14.2.A.3.3 | Mean TBI-223 Plasma Trough Concentrations by Treatment and Time Point, Approach to Steady State, Days 1 to 14<br>Cohort 3, PK Population |

### 14.2.B.1.1.1-14.2.B.1.3.2

## Individual Subjects TBI-223 Plasma Concentration by Treatment and Time Point, 0 to 24 Hours Post-dose

| 14.2.B.1.1.1 | Individual Subjects TBI-223 Plasma Concentration by Treatment and Time Point, Linear Scale Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state) Cohort 1, PK Population |
|---|---|
| 14.2.B.1.1.2 | Individual Subjects TBI-223 Plasma Concentration by Treatment and Time Point, Log-linear Scale Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state) Cohort 1, PK Population |

| 14.2.B.1.2.1 | Individual Subjects TBI-223 Plasma Concentration by Treatment and Time Point, Linear Scale Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state) Cohort 2, PK Population |
|---|---|
| 14.2.B.1.2.2 | Individual Subjects TBI-223 Plasma Concentration by Treatment and Time Point, Log-linear Scale Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state) Cohort 2, PK Population |
| 14.2.B.1.3.1 | Individual Subjects TBI-223 Plasma Concentration by Treatment and Time Point, Linear Scale<br>Hours 0 to 24 Post-Dose, Days 1 (single dose) and 14 (steady state)<br>Cohort 3, PK Population |
| 14.2.B.1.3.2 | Individual Subjects TBI-223 Plasma Concentration by Treatment and Time Point, Log-linear Scale Hours 0 to 24 Post-Dose, Days 1 (single dose) and 14 (steady state) Cohort 3, PK Population |

## 14.2.B.2.1.1-14.2.B.2.3.2

## Individual Subjects TBI-223 Plasma Concentration by Treatment and Time Point, 0 to 72 Hours Post-dose

| 14.2.B.2.1.1 | Individual Subjects TBI-223 Plasma Concentration by Treatment and Time Point, Linear Scale Hours 0 to 72 Post-Dose, Days 1 (single dose, fasted) and 17 (steady state, fed) Cohort 1, PK Population |
|---|---|
| 14.2.B.2.1.2 | Individual Subjects TBI-223 Plasma Concentration by Treatment and Time Point, Log-linear Scale Hours 0 to 72 Post-Dose, Days 1 (single dose, fasted) and 17 (steady state, fed) Cohort 1, PK Population |
| 14.2.B.2.2.1 | Individual Subjects TBI-223 Plasma Concentration by Treatment and Time Point, Linear Scale Hours 0 to 72 Post-Dose, Days 1 (single dose, fasted) and 17 (steady state, fed) Cohort 2, PK Population |
| 14.2.B.2.2.2 | Individual Subjects TBI-223 Plasma Concentration by Treatment and Time Point, Log-linear Scale Hours 0 to 72 Post-Dose, Days 1 (single dose, fasted) and 17 (steady state, fed) Cohort 2, PK Population |
| 14.2.B.2.3.1 | Individual Subjects TBI-223 Plasma Concentration by Treatment and Time Point, Linear Scale Hours 0 to 72 Post-Dose, Day 14 (steady state) Cohort 3, PK Population |

| Individual Subjects TBI-223 Plasma Concentration by Treatment and Time Point, Log-linear Scale | nours 0 to 72 Fost-Dose, Day 14 (steady state) Cohort 3, PK Population |
|---|---|
| 14.2.B.2.3.2 | |

### 14.2.B.3.1-14.2.B.3.3

# Individual Subjects TBI-223 Plasma Trough Concentration by Treatment and Time Point, Approach to Steady State

| 14.2.B.3.1 | Individual Subjects TBI-223 Plasma Trough Concentrations by Treatment and Time Point, Approach to Steady State, Days 4 to 17 Cohort 1, PK Population |
|---|---|
| 14.2.B.3.2 | Individual Subjects TBI-223 Plasma Trough Concentrations by Treatment and Time Point, Approach to Steady State, Days 4 to 17 Cohort 2, PK Population |
| 14.2.B.3.3 | Individual Subjects TBI-223 Plasma Trough Concentrations by Treatment and Time Point, Approach to Steady State, Days 1 to 14 Cohort 3, PK Population |

### 14.2.C.1.1.1-14.2.C.1.3.2

## Mean M2 Plasma Concentration by Treatment and Time Point, 0 to 24 Hours Post-dose

| 14.2.C.1.1.1 | Mean M2 Plasma Concentration by Treatment and Time Point, Linear Scale<br>Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state)<br>Cohort 1, PK Population |
|---|---|
| 14.2.C.1.1.2 | Mean M2 Plasma Concentration by Treatment and Time Point, Log-linear Scale<br>Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state)<br>Cohort 1, PK Population |
| 14.2.C.1.2.1 | Mean M2 Plasma Concentration by Treatment and Time Point, Linear Scale Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state) Cohort 2, PK Population |
| 14.2.C.1.2.2 | Mean M2 Plasma Concentration by Treatment and Time Point, Log-linear Scale<br>Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state)<br>Cohort 2, PK Population |
| 14.2.C.1.3.1 | Mean M2 Plasma Concentration by Treatment and Time Point, Linear Scale<br>Hours 0 to 24 Post-Dose, Days 1 (single dose) and 14 (steady state)<br>Cohort 3, PK Population |

| ule |
|---|
| Mean M2 Plasma Concentration by Treatment and Time Point, Log-linear Sci Hours 0 to 24 Post-Dose, Days 1 (single dose) and 14 (steady state) Cohort 3, PK Population |
| 14.2.C.1.3.2 |

### 14.2.C.2.1.1-14.2.C.2.3.2

## Mean M2 Plasma Concentration by Treatment and Time Point, 0 to 72 Hours Post-dose

| 14.2.C.2.1.1 | Mean M2 Plasma Concentration by Treatment and Time Point, Linear Scale<br>Hours 0 to 72 Post-Dose, Days 1 (single dose, fasted) and 17 (steady state, fed)<br>Cohort 1, PK Population |
|---|---|
| 14.2.C.2.1.2 | Mean M2 Plasma Concentration by Treatment and Time Point, Log-linear Scale<br>Hours 0 to 72 Post-Dose, Days 1 (single dose, fasted) and 17 (steady state, fed)<br>Cohort 1, PK Population |
| 14.2.C.2.2.1 | Mean M2 Plasma Concentration by Treatment and Time Point, Linear Scale<br>Hours 0 to 72 Post-Dose, Days 1 (single dose, fasted) and 17 (steady state, fed)<br>Cohort 2, PK Population |
| 14.2.C.2.2.2 | Mean M2 Plasma Concentration by Treatment and Time Point, Log-linear Scale<br>Hours 0 to 72 Post-Dose, Days 1 (single dose, fasted) and 17 (steady state, fed)<br>Cohort 2, PK Population |
| 14.2.C.2.3.1 | Mean M2 Plasma Concentration by Treatment and Time Point, Linear Scale<br>Hours 0 to 72 Post-Dose, Day 14 (steady state)<br>Cohort 3, PK Population |
| 14.2.C.2.3.2 | Mean M2 Plasma Concentration by Treatment and Time Point, Log-linear Scale<br>Hours 0 to 72 Post-Dose, Day 14 (steady state)<br>Cohort 3, PK Population |

### 14.2.C.3.1-14.2.C.3.3

## Mean M2 Plasma Trough Concentration by Treatment and Time Point, Approach to Steady State

| 14.2.C.3.1 | Mean M2 Plasma Trough Concentrations by Treatment and Time Point, Approach to Steady State, Days 4 to 17 |
|---|---|
| | Cohort 1, PK Population |

| 14.2.C.3.2 | Mean M2 Plasma Trough Concentrations by Treatment and Time Point, Approach to Steady State, Days 4 to 17 Cohort 2, PK Population |
|---|---|
| 14.2.C.3.3 | Mean M2 Plasma Trough Concentrations by Treatment and Time Point, Approach to Steady State, Days 1 to 14<br>Cohort 3, PK Population |

## 14.2.D.1.1.1-14.2.D.1.3.2

## Individual Subjects M2 Plasma Concentration by Treatment and Time Point, 0 to 24 Hours Post-dose

| 14.2.D.1.1.1 | Individual Subjects M2 Plasma Concentration by Treatment and Time Point, Linear Scale Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state) Cohort 1, PK Population |
|---|---|
| 14.2.D.1.1.2 | Individual Subjects M2 Plasma Concentration by Treatment and Time Point, Log-linear Scale<br>Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state)<br>Cohort 1, PK Population |
| 14.2.D.1.2.1 | Individual Subjects M2 Plasma Concentration by Treatment and Time Point, Linear Scale Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state) Cohort 2, PK Population |
| 14.2.D.1.2.2 | Individual Subjects M2 Plasma Concentration by Treatment and Time Point, Log-linear Scale Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state) Cohort 2, PK Population |
| 14.2.D.1.3.1 | Individual Subjects M2 Plasma Concentration by Treatment and Time Point, Linear Scale Hours 0 to 24 Post-Dose, Days 1 (single dose) and 14 (steady state) Cohort 3, PK Population |
| 14.2.D.1.3.2 | Individual Subjects M2 Plasma Concentration by Treatment and Time Point, Log-linear Scale<br>Hours 0 to 24 Post-Dose, Days 1 (single dose) and 14 (steady state)<br>Cohort 3, PK Population |

## 14.2.D.2.1.1-14.2.D.2.3.2

## Individual Subjects M2 Plasma Concentration by Treatment and Time Point, 0 to 72 Hours Post-dose

|--|--|

| 14.2.D.2.1.2 | Individual Subjects M2 Plasma Concentration by Treatment and Time Point, Log-linear Scale<br>Hours 0 to 72 Post-Dose, Days 1 (single dose, fasted) and 17 (steady state, fed)<br>Cohort 1, PK Population |
|---|---|
| 14.2.D.2.2.1 | Individual Subjects M2 Plasma Concentration by Treatment and Time Point, Linear Scale<br>Hours 0 to 72 Post-Dose, Days 1 (single dose, fasted) and 17 (steady state, fed)<br>Cohort 2, PK Population |
| 14.2.D.2.2.2 | Individual Subjects M2 Plasma Concentration by Treatment and Time Point, Log-linear Scale<br>Hours 0 to 72 Post-Dose, Days 1 (single dose, fasted) and 17 (steady state, fed)<br>Cohort 2, PK Population |
| 14.2.D.2.3.1 | Individual Subjects M2 Plasma Concentration by Treatment and Time Point, Linear Scale<br>Hours 0 to 72 Post-Dose, Day 14 (steady state)<br>Cohort 3, PK Population |
| 14.2.D.2.3.2 | Individual Subjects M2 Plasma Concentration by Treatment and Time Point, Log-linear Scale<br>Hours 0 to 72 Post-Dose, Day 14 (steady state)<br>Cohort 3, PK Population |

### 14.2.D.3.1-14.2.D.3.3

Individual Subjects M2 Plasma Trough Concentration by Treatment and Time Point, Approach to Steady State

| 14.2.D.3.1 | Individual Subjects M2 Plasma Trough Concentrations by Treatment and Time Point, Approach to Steady State, Days 4 to 17 Cohort 1, PK Population |
|---|---|
| 14.2.D.3.2 | Individual Subjects M2 Plasma Trough Concentrations by Treatment and Time Point, Approach to Steady State, Days 4 to 17 Cohort 2, PK Population |
| 14.2.D.3.3 | Individual Subjects M2 Plasma Trough Concentrations by Treatment and Time Point, Approach to Steady State, Days 1 to 14 Cohort 3, PK Population |

### Listings

| 16.1.7 | Subject Enrollment and Randomization |
|----------|--------------------------------------|
| 16.2.1.1 | Screen Failure |
| 16.2.1.2 | Subject Disposition |

Global Alliance for TB Drug Development Protocol No. TBI-223-CL-002 TKL No. P1980121

| 16.2.2 | Protocol Deviations |
|---|---|
| 16.2.3 | Population Datasets |
| 16.2.4.1 | Demographics and Baseline Characteristics |
| 16.2.4.2 | Prior and Concomitant Medication |
| 16.2.4.3 | Medical and Surgical History |
| 16.2.5.1 | Plasma Concentration Values |
| 16.2.5.2 | TBI-223 Pharmacokinetic Parameters |
| 16.2.5.3 | TBI-223 Elimination Rate Constant and Half-Life |
| 16.2.5.4 | M2 Pharmacokinetic Parameters |
| 16.2.5.5 | M2 Elimination Rate Constant and Half-Life |
| 16.2.5.6 | Fasting and Meals |
| 16.2.7.1 | Adverse Events |
| 16.2.7.2 | Serious Adverse Events and Adverse Events Leading to Study Discontinuation |
| 16.2.8.1 | Childbearing Potential and Serum Pregnancy Tests |
| 16.2.8.2 | Urine Drug Screen and Alcohol Screenings |
| 16.2.8.3 | Clinical Laboratory Tests – Investigator's Assessments |
| 16.2.8.4.1 | Clinical Laboratory Test Results: Serum Chemistry |
| 16.2.8.4.2 | Clinical Laboratory Test Results: Hematology |
| 16.2.8.4.3 | Clinical Laboratory Test Results: Urinalysis |
| 16.2.8.4.4 | Clinical Laboratory Test Results: Coagulation |
| 16.2.8.5 | Laboratory Values Outside of Normal Range |
| 16.2.8.6 | Vital Signs |
| 16.2.8.7.1 | Physical Examinations |
| 16.2.8.7.2 | Neurological Examinations |
| 16.2.8.8 | 12-Lead ECG Results |
| 16.2.9 | General Comments |


Table 14.1.1: Summary of Subject Disposition

| | TBI-223<br>1800 mg | TBI-223<br>2400 mg | TBI-223<br>3000 mg | Any TBI-223 | Pooled Placebo | Overall |
|---|---|---|---|---|---|---|
| Number of Subjects Screened | | | | | | XX |
| Number of Subjects Randomized | XX | X | XX | XX | XX | XX |
| Number of Subjects in Safety Population, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| (PK) Population, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Number of Subjects Completing the Study, | (X XX) XX | (X XX) XX | (A AA) AA | | (X XX) XX | (X XX) XX |
| Number of Subjects Discontinued, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Keason for Discontinuation, n (70)<br>Withdrawal of Informed Consent | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Adverse Event/Serious Adverse Event | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Subject's Request | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| Protocol Violation | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Occurrence of one of the safety criteria for exclusion after treatment has been instituted | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XXX)XX | (XXX)XX | (XXXX) |
| Subject is Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Investigator's Judgment | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other[1] | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Denominator for percentages is the number of subjects randomized.

[1] See subject comment for details. <Programming Note: Include this footnote only if applicable. If multiple subjects have the same reason specified as a comment, include a row for that reason.>

Generated on XX/XX/XXXXXX by XXXXX / Uses: XXXX / Reference: Data Listing XXXX

Page X of Y

Table 14.1.2: Summary of Subject Demographics and Baseline Characteristics Safety Population

| | TBI-223<br>1800 mg | TBI-223<br>2400 mg | TBI-223<br>3000 mg | Any TBI-223 | Pooled Placebo | Overall |
|---|---|---|---|---|---|---|
| Age (years) Mean (SD) Median Minimum, Maximum | XX.XX (XX.XX)<br>XX.X<br>XX.X, XX.X | XX.XX (XX.XX)<br>XX.X<br>XX.X, XX.X | XX.XX (XX.XX)<br>XX.X<br>XX.X, XX.X | XX.XX (XX.XX)<br>XX.X<br>XX.X, XX.X | XX.XX (XX.XX)<br>XX.X<br>XX.X, XX.X | XX.XX (XX.XX)<br>XX.X<br>XX.X, XX.X |
| Gender, n (%)<br>Male<br>Female | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| Race, n (%) White Black or African | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| American<br>Asian<br>American Indian | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| or Alaskan Native<br>Native Hawaiian<br>or Other Pacific | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Islander<br>Other/Multiracial | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Page X of Y

Table 14.1.2: Summary of Subject Demographics and Baseline Characteristics Safety Population

| | TBI-223<br>1800 mg | TBI-223<br>2400 mg | TBI-223<br>3000 mg | Any TBI-223 | Pooled Placebo | Overall |
|---|---|---|---|---|---|---|
| Ethnicity, n(%) Hispanic or Latino Not Hispanic or Latino | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Weight (kg) Mean (SD) Median Minimum, Maximum | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Height (cm) Mean (SD) Median Minimum, Maximum | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) | XX.XX (XX.XX) |
| | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| BMI (kg/m², [1]<br>Mean (SD)<br>Median<br>Minimum,<br>Maximum | XX.XX (XX.XX)<br>XX.X<br>XX.X, XX.X | XX.XX (XX.XX)<br>XX.X<br>XX.X, XX.X | XX.XX (XX.XX)<br>XX.X<br>XX.X, XX.X | XX.XX (XX.XX)<br>XX.X<br>XX.X, XX.X | XX.XX (XX.XX)<br>XX.X<br>XX.X, XX.X | XX.XX (XX.XX)<br>XX.X<br>XX.X, XX.X |

[1] Baseline BMI is calculated as baseline weight / baseline height^2.

Generated on XX/XX/XX:XXXX by XXXX / Uses: XXXX / Reference: Data Listing XXXX


Page X of Y

Table 14.1.3.1: Summary of Extent of Exposure of TBI-223
Safety Population

| | for Cohort 1 (1800<br>mg)/Cohort 2 (2400<br>mg) | Study Day of Dose<br>for Cohort 3 (3000<br>mg) | 1800 mg<br>(N=XX) | 1B1-223<br>2400 mg<br>(N=XX) | 1B1-223<br>3000 mg<br>(N=XX) | Any 1B1-223<br>(N=XX) |
|---|---|---|---|---|---|---|
| Subjects who Received Treatment, N (%) | | | | | | |
| At Least One Dose | | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| All Intended Doses | 15 total | 14 total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Fasting Dose | Day 1 | | XX (XX.X) | XX (XX.X) | ł | XX (XX.X) |
| Fed Doses | | | | | | |
| Dose 1 | Day 4 | Day 1 | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| Dose 2 | Day 5 | Day 2 | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) |
| Dose 3 | Day 6 | Day 3 | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| Dose 4 | Day 7 | Day 4 | XX(XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) |
| Dose 5 | Day 8 | Day 5 | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) |
| Dose 6 | Day 9 | Day 6 | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) |
| Dose 7 | Day 10 | Day 7 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| Dose 8 | Day 11 | Day 8 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| Dose 9 | Day 12 | Day 9 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| Dose 10 | Day 13 | Day 10 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| Dose 11 | Day 14 | Day 11 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| Dose 12 | Day 15 | Day 12 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| Dose 13 | Day 16 | Day 13 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| Dose 14 | Day 17 | Day 14 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total Number of Doses | | | | | | |
| Z | | | XX | XX | XX | XX |
| Mean (SD) | | | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | | | XXX.X | XXX.X | XX.X | XXX.X |
| Minimum, Maximum | | | XX, XX | XX, XX | XX, XX | XX, XX |

Generated on XX/XX/XX:XXXX by XXXX / Uses: XXXX / Reference: Data Listing XXXX


Page X of Y

Table 14.2.1.X: Summary of Plasma TBI-223 Concentration (ng/mL) by Time Point [TBI-223 1800mg] [TBI-223 2400mg] [TBI-223 3000mg]

Pharmacokinetic (PK) Population

| | | | L | TBI-223 | | | | | | M2 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Z | N Mean (SD) | Geometric<br>Mean (SE) | CV (%) | Minimum,<br>Maximum | Median | Z | Mean (SD) | Geometric<br>Mean (SE) | CV (%) | Minimum,<br>Maximum | Median |
| Day 1 | | | | | | | | | | | | |
| Pre-Dose | XX | xxx (xxx) | (xxx (xxx) | XX.X | XXX, XXX | XXX | XX | xxx (xxx) | xxx (xxx) | XX.X | XXX, XXX | XXX |
| 30 Minutes | XX | (xxx) xxx | (xxx) xxx | x.x.x | xxx, xxx | xxx | XX | (xxx) xxx | (xxx) xxx | x.x.x | xxx, xxx | xxx |
| 1 Hour | XX | (xxx) xxx | (xxx) xxx | x.xx | xxx, xxx | XXX | XX | xxx (xxx) | (xxx) xxx | XX.X | xxx, xxx | xxx |
| 2 Hours | XX | (xxx) xxx | (xxx) xxx | x.xx | xxx, xxx | XXX | XX | xxx (xxx) | (xxx) xxx | XX.X | xxx, xxx | xxx |
| 3 Hours | XX | (xxx) xxx | (xxx) xxx | XX.X | xxx, xxx | XXX | XX | (xxx) xxx | (xxx) xxx | XX.X | xxx, xxx | xxx |
| 4 Hours | XX | xxx (xxx) | (xxx) xxx | XX.X | XXX, XXX | XXX | XX | xxx (xxx) | (xxx) xxx | XX.X | XXX, XXX | XXX |
| 5 Hours | XX | (xxx) xxx | (xxx) xxx | XX.X | XXX, XXX | XXX | XX | xxx (xxx) | (xxx) xxx | X.X.X | XXX, XXX | XXX |
| 6 Hours | XX | xxx(xxx) | (xxx) xxx | xx.x | xxx, xxx | XXX | XX | xxx (xxx) | (xxx) xxx | X.X.X | xxx, xxx | XXX |
| 7 Hours | XX | (xxx) xxx | (xxx) xxx | xx.x | xxx, xxx | XXX | XX | xxx (xxx) | (xxx) xxx | XX.X | xxx, xxx | XXX |
| 8 Hours | XX | (xxx) xxx | (xxx) xxx | x.xx | xxx, xxx | XXX | XX | xxx (xxx) | (xxx) xxx | XX.X | xxx, xxx | xxx |
| 12 Hours | XX | (xxx) xxx | (xxx) xxx | x.xx | xxx, xxx | XXX | XX | xxx (xxx) | (xxx) xxx | XX.X | xxx, xxx | xxx |
| 16 Hours | XX | (xxx) xxx | (xxx) xxx | xx.x | xxx, xxx | xxx | XX | xxx (xxx) | (xxx) xxx | x.xx | xxx, xxx | XXX |
| 20 Hours | XX | xxx (xxx) | (xxx) xxx | XX.X | XXX, XXX | XXX | XX | xxx (xxx) | (xxx) xxx | XX.X | XXX, XXX | XXX |
| 24 Hours | XX | (xxx) xxx | (xxx) xxx | XX.X | xxx, xxx | XXX | XX | xxx (xxx) | (xxx) xxx | XX.X | xxx, xxx | xxx |
| 30 Hours | XX | (xxx) xxx | (xxx) xxx | xx.x | xxx, xxx | XXX | XX | xxx (xxx) | (xxx) xxx | XX.X | xxx, xxx | XXX |
| 36 Hours | XX | (xxx) xxx | (xxx) xxx | XX.X | xxx, xxx | XXX | XX | xxx (xxx) | (xxx) xxx | XX.X | xxx, xxx | xxx |
| <etc.></etc.> | | | | | | | | | | | | |

Note: Concentrations below the limit of quantitation are imputed as 0.00 in the computation of descriptive statistics. SD = Standard Deviation, SE = Standard Error, CV Coefficient of Variation.

Generated on XX/XX/XX:XXXX by XXXXX / Uses: XXXX / Reference: Data Listing XXXX

Note: Include all measured time points for all cohorts. Label pre-dose time points for Days 5-17 (Cohorts 1 and 2) and Days 2-14(Cohort 3) as Crough (pre-dose).


Table 14.2.2.1.X: Summary of TBI-223 Pharmacokinetic Parameters [TBI-223 1800mg] [TBI-223 2400mg] Pharmacokinetic (PK) Population

| | | | Da | ay 1 (fasting) | | | | | D | Day 4 (fed) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Z | Geometric N Mean (SD) Mean (SE) | Geometric<br>Mean (SE) | (%) A) | Minimum,<br>Maximum | Median | Z | Mean (SD) | Geometric Median N Mean (SD) Mean (SE) | (%) | Minimum,<br>Maximum | Median |
| | ; | (20) | (22) | (2.) | | | ; | | (76) | (a) | | |
| $AUC_{0.24} (\mu g^*h/mL)$ xx xxx (xxx) | X | (xxx) xxx | (xxx) xxx | XX.X | XXX, XXX | XXX | XX | (xxx (xxx) | (xxx) xxx | X.X.X | XXX, XXX | XXX |
| $\mathrm{AUC}_{\mathrm{inf}}\left(\mu g^{*}h/\mathrm{mL}\right)$ | XX | xxx (xxx) | (xxx) xxx | XX.X | XXX, XXX | XXX | XX | (xxx) xxx | (xxx) xxx | XX.X | xxx, xxx | XXX |
| $C_{max} (\mu g/mL)$ | XX | xxx (xxx) | (xxx) xxx | XX.X | xxx, xxx | XXX | XX | (xxx) xxx | (xxx) xxx | X.X.X | xxx, xxx | XXX |
| $T_{max}(h)$ | XX | xxx (xxx) | 1 | 1 | xxx, xxx | XXX | XX | (xxx) xxx | 1 | ŀ | xxx, xxx | XXX |
| $\lambda_{\mathrm{z}}$ (/h) | XX | xxx (xxx) | 1 | 1 | xxx, xxx | XXX | XX | (xxx) xxx | 1 | 1 | xxx, xxx | XXX |
| $\mathfrak{t}_{2}\left(\mathrm{h}\right)$ | XX | xxx (xxx) | 1 | ŀ | xxx, xxx | XXX | XX | (xxx) xxx | : | 1 | XXX, XXX | XXX |
| CL/F (L/h) | XX | xxx (xxx) | 1 | 1 | XXX, XXX | XXX | XX | (xxx) xxx | 1 | ŀ | xxx, xxx | XXX |
| $V_Z/F$ (L) | XX | (xxx) xxx xx | 1 | 1 | xxx, xxx | XXX | XX | (xxx) xxx | 1 | ! | xxx, xxx | XXX |

Note: Concentrations below the limit of quantitation are imputed as 0 in the computation of  $AUC_{0-24}$ . SD = Standard Deviation, SE = Standard Error, CV = Coefficient of Variation.

Generated on XX/XX/XX:XXXX by XXXXX / Uses: XXXX / Reference: Data Listing XXXX


Table 14.2.2.2.X: Summary of TBI-223 Pharmacokinetic Parameters [TBI-223 1800mg] [TBI-223 2400mg] [All Subjects] [Male Subjects] Pharmacokinetic (PK) Population

| | N | Mean (SD) | Geometric Mean (SE) | CV (%) | CV (%) Minimum, Maximum | Median |
|---|---|---|---|---|---|---|
| Day 4 (fed, single-dose) | | | | | | |
| $AUC_{0-24}$ ( $\mu g*h/mL$ ) | XX | (xxx) xxx | xxx (xxx) | x.x.x | XXX, XXX | xxx |
| $AUC_{inf}(\mu g^*h/mL)$ | XX | xxx(xxx) | xxx (xxx) | x.x.x | xxx, xxx | xxx |
| $C_{max}$ ( $\mu g/mL$ ) | XX | xxx(xxx) | xxx (xxx) | x.xx | XXX, XXX | XXX |
| $T_{max}$ (h) | XX | (xxx) xxx | 1 | ; | XXX, XXX | xxx |
| $\lambda_{z}$ (/h) | XX | xxx(xxx) | 1 | ; | XXX, XXX | xxx |
| $\mathrm{t}_{\flat_2}(\mathrm{h})$ | XX | xxx (xxx) | : | 1 | XXX, XXX | XXX |
| Day 17 (fed, steady state) | | | | | | |
| $AUC_{0-24}$ ( $\mu g*h/mL$ ) | XX | (xxx) xxx | xxx (xxx) | x.x.x | XXX, XXX | xxx |
| $AUC_{inf}(\mu g^*h/mL)$ | XX | (xxx) xxx | (XXX (XXX) | X.X.X | XXX, XXX | xxx |
| $\mathrm{C}_{\mathrm{max}}\left(\mu\mathrm{g/mL} ight)$ | XX | (xxx) xxx | xxx (xxx) | x.xx | XXX, XXX | xxx |
| $T_{ m max} \left( { m h} ight)$ | XX | (xxx) xxx | 1 | 1 | XXX, XXX | xxx |
| $C_{min}$ ( $\mu g/mL$ ) | XX | (xxx) xxx | 1 | 1 | XXX, XXX | xxx |
| $T_{min}\left(h\right)$ | XX | (xxx) xxx | 1 | 1 | XXX, XXX | xxx |
| $\lambda_{\mathrm{z}}\left(/\mathrm{h}\right)$ | XX | (xxx) xxx | : | ; | XXX, XXX | xxx |
| t <sub>2</sub> , (h) | XX | xxx (xxx) | ; | 1 | XXX, XXX | XXX |
| Accumulation Ratio | | | | | | |
| C <sub>max</sub> | XX | (xxx (xxx) | : | ; | XXX, XXX | XXX |
| $\mathrm{AUC}_{0-24}$ | XX | (xxx) xxx | : | ; | XXX, XXX | XXX |

Note: Concentrations below the limit of quantitation are imputed as 0 in the computation of AUC<sub>0-24</sub>. SD = Standard Deviation, SE = Standard Error, CV = Coefficient of Variation.

Generated on XX/XX/XX:XXXX by SMYXX / Uses: XXXX / Reference: Data Listing XXXX


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002

Table 14.2.2.2.3: Summary of TBI-223 Pharmacokinetic Parameters TBI-223 3000mg [All Subjects][Male Subjects][Female Subjects] Pharmacokinetic (PK) Population

| | Z | Mean (SD) | Geometric Mean (SE) | CV (%) | Minimum,<br>Maximum | Median |
|---|---|---|---|---|---|---|
| Day 1 (fed, single-dose) | | | | | | |
| $^{\star}$ AUC <sub>0-24</sub> ( $\mu g^*h/mL$ ) | XX | (xxx (xxx) | (XXX (XXX) | XX.X | XXX, XXX | XXX |
| AUCinf (µg*h/mL) | XX | xxx(xxx) | (XXX)(XXX) | XX.X | XXX, XXX | XXX |
| $C_{max}$ ( $\mu g/mL$ ) | XX | xxx(xxx) | (xxx)(xxx) | XX.X | XXX, XXX | XXX |
| $T_{\mathrm{max}}\left(\mathrm{h}\right)$ | XX | xxx(xxx) | I | 1 | XXX, XXX | XXX |
| $\lambda_{ m z}\left(/{ m h} ight)$ | XX | xxx(xxx) | ŀ | 1 | XXX, XXX | XXX |
| t <sub>2</sub> , (h) | XX | xxx(xxx) | I | 1 | XXX, XXX | XXX |
| CL/F $(L/h)$ | XX | xxx(xxx) | 1 | 1 | XXX, XXX | XXX |
| $ m V_Z/F~(L)$ | XX | (xxx) xxx | ŀ | 1 | XXX, XXX | XXX |
| Day 14 (fed, steady state) | | | | | | |
| $AUC_{0-24}$ ( $\mu g*h/mL$ ) | XX | xxx(xxx) | (xxx)(xxx) | XX.X | XXX, XXX | XXX |
| $AUC_{inf}(\mu g^*h/mL)$ | XX | xxx(xxx) | (xxx)xxx | XX.X | XXX, XXX | XXX |
| $C_{max}$ ( $\mu g/mL$ ) | XX | xxx(xxx) | (xxx)xxx | XX.X | XXX, XXX | XXX |
| $T_{ m max} \left( m h ight)$ | XX | xxx(xxx) | 1 | 1 | XXX, XXX | XXX |
| Cmin (µg/mL) | XX | xxx(xxx) | ı | 1 | XXX, XXX | XXX |
| $T_{min}$ (h) | XX | xxx(xxx) | ! | 1 | XXX, XXX | XXX |
| $\lambda_{\mathrm{z}}\left(/\mathrm{h} ight)$ | XX | (xxx) xxx | ŀ | 1 | xxx, xxx | XXX |
| $\mathbf{t}_{\lambda_{2}}(\mathbf{h})$ | XX | (xxx) xxx | : | ŀ | XXX, XXX | XXX |
| Accumulation Ratio | | | | | | |
| Cmax | XX | (xxx) xxx | (XXX (XXX) | XX.X | XXX, XXX | XXX |
| $\mathrm{AUC}_{0.24}$ | XX | (xxx) xxx | (xxx) xxx | XX.X | XXX, XXX | XXX |

Note: Concentrations below the limit of quantitation are imputed as 0.00 in the computation of AUC<sub>0-24</sub>. SD = Standard Deviation, SE = Standard Error, CV = Coefficient of Variation.

Generated on XX/XX/XX:XXXX by SMYXX / Uses: XXXX / Reference: Data Listing XXXX

Global Alliance for TB Drug Development Protocol No. TBI-223-CL-002 TKL No. P1980121 Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002


## Table 14.2.3: Summary of TBI-223 Pharmacokinetic Parameters Food Effect Pharmacokinetic (PK) Population

| | TBI-223 1800 mg (N=xx) | TBI-223 2400mg (N=xx) |
|---|---|---|
| C <sub>max</sub> (μg/mL) Fasting Geometric Mean (SEM) Fed Geometric Mean (SEM) Ratio of Geometric Means 90% Confidence Interval | X.XXX (X.XXX) X.XXX (X.XXX) X.XXX [X.XXX] | x.xxx (x.xxx)<br>x.xxx (x.xxx)<br>x.xxx<br>[x.xxx, x.xxx] |
| AUC₀-24 (μg.h/mL) Fasting Geometric Mean (SEM) Fed Geometric Mean (SEM) Ratio of Geometric Means 90% Confidence Interval | X.XXX (X.XXX) X.XXX (X.XXX) X.XXX [X.XXX] | x.xxx (x.xxx)<br>x.xxx (x.xxx)<br>x.xxx<br>[x.xxx, x.xxx] |
| AUC <sub>inf</sub> (μg.h/mL) Fasting Geometric Mean (SEM) Fed Geometric Mean (SEM) Ratio of Geometric Means 90% Confidence Interval | x.xxx (x.xxx)<br>x.xxx (x.xxx)<br>x.xxx<br>[x.xxx, x.xxx] | x.xxx (x.xxx)<br>x.xxx (x.xxx)<br>x.xxx<br>[x.xxx, x.xxx] |
| T <sub>max</sub> (h) Fasting Median Fed Median P value (Wilcoxon Signed Rank test, Fed vs. Fasting) | X.XX<br>X.XX<br>X.XXX | X.XX<br>X.XX<br>X.XXX |

Note: Generated on XX/XX/XX:XXXX by SMYXX / Uses: XXXX / Reference: Data Listing XXXX


Table 14.2.4: Summary of TBI-223 Pharmacokinetic Parameters Confirmation of Steady State Pharmacokinetic (PK) Population

| TBI-223 3000mg $(N=xx)$ | X.XXX<br>X.XXX |
|---|---|
| TBI-223 2400mg $(N=xx)$ | X.XXX<br>X.XXX |
| TBI-223 1800 mg (N=xx) | X.XXX<br>X.XXX |
| | P value (study day; slope)<br>P value (subject-day interaction) |

Note: For 1800mg and 2400mg, the analysis includes pre-dose concentrations for Days 10 through 17, and 24h concentration for Day 17; for 3000mg, the analysis includes pre-dose concentrations for Days 7 through 14, and 24h concentration for Day 14.

Generated on XX/XX/XX:XXXX by SMYXX / Uses: XXXX / Reference: Data Listing XXXX


Table 14.2.5: Summary of TBI-223 Pharmacokinetic Parameters Analysis of Gender Differences Pharmacokinetic (PK) Population

| | TBI-223 | TBI-223 1800 mg | TBI-223 | TBI-223 2400mg | TBI-223 | TBI-223 3000mg |
|---|---|---|---|---|---|---|
| | Male | Female | Male | Female | Male | Female |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| , , , | | | | | | |
| Single-Dose, Fed[a] | | | | | | |
| Cmax (µg/mL) | | | | | | |
| Arithmetic Mean (SD) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX (X.XXX) | X.XXX (X.XXX) X.XXX (X.XXX) X.XXX (X.XXX) | X.XXX (X.XXX) | X.XXX (X.XXX) |
| Geometric Mean (SEM) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX (X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) |
| P value (gender, t test) | | X.XXX | | X.XXX | | X.XXX |
| AUC <sub>0-24</sub> (µg.h/mL) | | | | | | |
| Arithmetic Mean (SD) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) |
| Geometric Mean (SEM) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) | | X.XXX(X.XXX) | X.XXX(X.XXX) |
| P value (gender, $t$ test) | | X.XXX | | X.XXX | | X.XXX |

[a] Day 4 for 1800mg and 2400mg, Day 1 for 3000mg.


Table 14.2.5: Summary of TBI-223 Pharmacokinetic Parameters Analysis of Gender Differences Pharmacokinetic (PK) Population

| | TBI-223 | TBI-223 1800 mg | TBI-223 | TBI-223 2400mg | TBI-223 | TBI-223 3000mg |
|---|---|---|---|---|---|---|
| | Male (N=xx) | Female (N=xx) | Male (N=xx) | Female (N=xx) | Male (N=xx) | Female (N=xx) |
| Steady State, Fed[a] | | | | | | |
| С <sub>max</sub> (µg/mL) | | | | | | |
| Arithmetic Mean (SD) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) |
| Geometric Mean (SEM) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) |
| P value (gender, $t$ test) | | X.XXX | | X.XXX | | X.XXX |
| AUC <sub>0-24</sub> (μg.h/mL) | | | | | | |
| Arithmetic Mean (SD) | X.XXX(X.XXX) | X.XXX (X.XXX) | X.XXX (X.XXX) | | X.XXX (X.XXX) X.XXX (X.XXX) | X.XXX (X.XXX) |
| Geometric Mean (SEM) | X.XXX(X.XXX) | X.XXX(X.XXX) | | X.XXX(X.XXX) | x.xxx(x.xxx) | x.xxx(x.xxx) |
| P value (gender, t test) | | X.XXX | | X.XXX | | X.XXX |

[a] Day 17 for 1800mg and 2400mg, Day 14 for 3000mg.


Table 14.2.5: Summary of TBI-223 Pharmacokinetic Parameters Analysis of Gender Differences Pharmacokinetic (PK) Population

| | TBI-223 | TBI-223 1800 mg | TBI-223 | TBI-223 2400mg |
|---|---|---|---|---|
| | Male | Female | Male | Female |
| | (XX=N) | (XX=NI) | (XX=N) | (XX=N) |
| Single Dose, Fasting (Day 1) | | | | |
| C <sub>max</sub> (µg/mL) | | | | |
| Arithmetic Mean (SD) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) |
| Geometric Mean (SEM) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) |
| P value (gender, $t$ test) | | X.XXX | | X.XXX |
| AUC <sub>0-24</sub> (μg.h/mL) | | | | |
| Arithmetic Mean (SD) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) | X.XXX(X.XXX) |
| Geometric Mean (SEM) | X.XXX(X.XXX) | X.XXX(X.XXX) | x.xxx(x.xxx) | X.XXX(X.XXX) |
| P value (gender, $t$ test) | | X.XXX | | X.XXX |

Note: Tables 14.2.6.1.1 through 14.2.9 follow identical layouts to 14.2.2.1.1 through 14.2.5.

Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002

| | TBI-223 | TBI-223 | TBI-223 | Any | Pooled |
|---|---|---|---|---|---|
| | 1800 mg | 2400 mg | 3000 mg | TBI-223 | Placebo |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Treatment-Emergent Adverse Events (TEAEs) Number of Events Number of Subjects, n (%) | XX | XX | XX | XX | XX |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Treatment-Related TEAEs<br>Number of Events<br>Number of Subjects, n (%) | XX<br>XX (XX.X) | XX<br>XX (XX.X) | XX<br>XX (XXX.X) | XX<br>XX (XX.X) | XX<br>XX (XX.X) |
| Serious TEAEs (All) Number of Events Number of Subjects, n (%) | XX | XX | XX | XX | XX |
| | XX (XX.X) | XX (XX.X) | XX (XXX.X) | XX (XX.X) | XX (XX.X) |
| Serious TEAEs (Deaths) Number of Events Number of Subjects, n (%) | XX | XX | XX | XX | XX |
| | XX (XX.X) | XX (XX.X) | XX (XXX.X) | XX (XX.X) | XX (XX.X) |
| Treatment-Related Serious TEAEs Number of Events Number of Subjects, n (%) | XX | XX | XX | XX | XX |
| | XX (XX.X) | XX (XX.X) | XX (XXX.X) | XX (XX.X) | XX (XX.X) |
| TEAEs Leading to Study Discontinuation Number of Events Number of Subjects, n (%) | XX | XX | XX | XX | XX |
| | XX (XX.X) | XX (XX.X) | XX (XXX.X) | XX (XX.X) | XX (XX.X) |

Note: TEAEs include all AEs starting or worsening after the first dosing of the study drug.


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002

Page X of Y

Table 14.3.1.2: Summary of Treatment-Emergent Adverse Events by Preferred Term in Descending Frequency Safety Population

| | TBI-223<br>1800 mg<br>(N=XX) | TBI-223<br>2400 mg<br>(N=XX) | TBI-223<br>3000 mg<br>(N=XX) | Any<br>TBI-223<br>(N=XX) | Pooled Placebo (N=XX) |
|---|---|---|---|---|---|
| Subjects with Any TEAE, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| < <adverse event="" preferred="" term="">&gt; &lt;<adverse event="" preferred="" term="">&gt;</adverse></adverse> | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |

Note: TEAEs include all AEs starting or worsening on or after the dosing of the study drug. Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA preferred term. Each subject will be counted only once within a preferred term.

Generated on XX/XX/XX:XXXX by XXXX / Uses: XXXX / Reference: Data Listing XXXX

[Programming note: AEs will be presented in descending order of the frequency of PT in the "Any-TBI-223" column.]

Page X of Y

Table 14.3.1.3: Summary of Treatment-Related Treatment-Emergent Adverse Events by Preferred Term in Descending Frequency Safety Population

| | TBI-223<br>1800 mg<br>(N=XX) | TBI-223<br>2400 mg<br>(N=XX) | TBI-223<br>3000 mg<br>(N=XX) | Any<br>TBI-223<br>(N=XX) | Pooled Placebo<br>(N=XX) |
|---|---|---|---|---|---|
| Subjects with Any Treatment-Related TEAE, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| < <adverse event="" preferred="" term="">&gt; &lt;<adverse event="" preferred="" term="">&gt;</adverse></adverse> | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |

Note: TEAEs include all AEs starting or worsening on or after the dosing of the study drug. Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA preferred term. Each subject will be counted only once within a preferred term.

Generated on XX/XX/XX:XXXX by XXXX / Uses: XXXX / Reference: Data Listing XXXX

[Programming note: AEs will be presented in descending order of the frequency of PT in the "Any-TBI-223" column.]


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002

r: 1BI-223-CL-002 Table 14.3.1.4: Summary of Treatn

Table 14.3.1.4: Summary of Treatment-emergent Adverse Events by System Organ Class and Preferred Term by Maximum Severity Safety Population

| | TBI-223<br>1800 mg | TBI-223<br>2400 mg | TBI-223<br>3000 mg | Any<br>TBI-223 | Pooled Placebo |
|---|---|---|---|---|---|
| | (XXX ) (1) | (XXX ) (1) | (*** ) | (XXXZ_11) | (**** |
| Subjects with Any TEAE, n (%) | | | | | |
| Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Mild | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| Severe | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Potentially Life-Threatening | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| << Adverse Fvent Body System>> | | | | | |
| Harden Doug by Stome | | | | | |
| lotal | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX (XX.X) |
| Mild | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| Potentially Life-Threatening | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| < <adverse event="" preferred="" term="">&gt;</adverse> | | | | | |
| Total | XX(XX.X) | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| Mild | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX (XX.X) |
| Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| Potentially Life-Threatening | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: TEAEs include all AEs starting or worsening on or after the dosing of the study drug. Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA preferred term. Each subject will be counted only once within a system organ class or a preferred term.

Generated on XX/XX/XX:XXXX by XXXX / Uses: XXXX / Reference: Data Listing XXXX

[Programming note: AEs will be presented in alphabetical order of SOC and descending order by the descending frequency of PT in the "Any TBI-223" column]

Page X of Y

Table 14.3.1.5: Summary of Treatment-Related Treatment-emergent Adverse Events by System Organ Class and Preferred Term by Maximum Severity Safety Population

| | TBI-223<br>1800 mg<br>(N=XX) | TBI-223<br>2400 mg<br>(N=XX) | TBI-223<br>3000 mg<br>(N=XX) | Any<br>TBI-223<br>(N=XX) | Pooled Placebo (N=XX) |
|---|---|---|---|---|---|
| Subjects with Any Treatment-Related TEAE, n (%) Total Mild Moderate Severe Potentially Life-Threatening | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <pre>&lt;&lt; Adverse Event Body System&gt;&gt;</pre> | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) |
| <>Adverse Event Preferred Term>> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: TEAEs include all AEs starting or worsening on or after the dosing of the study drug. Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA preferred term. Each subject will be counted only once within a system organ class or a preferred term.


Page X of Y

Table 14.3.1.6: Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term by Maximum Causality Safety Population

| | TBI-223 | TBI-223 | TBI-223 | Any | Pooled |
|---|---|---|---|---|---|
| | 1800 mg (N=XX) | 2400 mg $(N=XX)$ | 3000 mg<br>(N=XX) | TBI-223 (N=XX) | Placebo<br>(N=XX) |
| Subjects with Any TEAE, n (%) | | | | | |
| Total | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| Not Related | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| Unlikely | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| Possible | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| Probable | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| Certain | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Body System>> | | | | | |
| Total | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Related | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Unlikely | XX(XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Possible | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Probable | XX(XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Certain | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| < <adverse event="" preferred="" term="">&gt;</adverse> | | | | | |
| Total | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| Not Related | XX(XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Unlikely | XX(XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Possible | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Probable | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Certain | XX(XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: TEAEs include all AEs starting or worsening on or after the dosing of the study drug. Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA preferred term. Each subject will be counted only once within a system organ class or a preferred term.

Global Alliance for TB Drug Development

Protocol Number: TBI-223-CL-002

Table 14.3.2.1.X: Summary of Clinical [Hematology][ Chemistry][Coagulation] Absolute Values and Change from Baseline by Treatment and Time Point Safety Population

| | TBI-223<br>1800 mg<br>(N=XX) | TBI-223<br>2400 mg<br>(N=XX) | TBI-223<br>3000 mg<br>(N=XX) | Pooled<br>Placebo<br>(N=XX) |
|---|---|---|---|---|
| [Lab Tests Name (Units)] Day -1 (Baseline) N | XX | ** | × | XX |
| Mean (SD)<br>Median | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX | XX, XX |
| Day 1, 6-7 hours post-dose | XX | ×× | ×× | XX |
| Mean (SD)<br>Median | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX | XX, XX |
| Change from Baseline<br>N | XX | XX | XX | XX |
| Mean (SD)<br>Median<br>Minimum, Maximum | XX.X (XX.X)<br>XX<br>XX, XX | XX.X (XX.X)<br>XX<br>XX, XX | XX.X (XX.X)<br>XX<br>XX, XX | XX.X (XX.X)<br>XX<br>XX, XX |

Note: Baseline is the last available measurement prior to the first dose of the study drug on Day 1. If Day -1 Assessment is missing, use Screening Assessment. Generated on XX/XX/XX:XXXX by XXX / Uses: XXXX / Reference: Data Listing XXXX Continue for safety labs (hematology and chemistry) and Coagulation at 6-7 hours post-dose on Days 1, 2, 3, 4, 6, 10, 14, 17, and on Days 20 and 26

[Programming Note: Summarize all lab tests with continuous results. Page break between lab tests.]

Page X of Y

Table 14.3.2.2.X: Summary of Clinical [Hematology][ Chemistry][Coagulation] Categorical Change from Baseline

Safety Population

| [Lab Tests Name (Units)] Day 1 Number of Subjects Assessed, N (%) Below Normal -> Below Normal Below Normal -> Above Normal XX.X (XX.X) XX.X (XX.X) Below Normal -> Above Normal Normal -> Below Normal XX.X (XX.X) | XX | | (N=XX) | (X=X) |
|---|---|---|---|---|
| | XX | | | |
| | | XX | XX | XX |
| | .X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X(XX.X) |
| Normal -> Normal XX.X (XX.X) | .X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X(XX.X) |
| Normal -> Above Normal XX.X (XX.X) | .X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X(XX.X) |
| Above Normal -> Below Normal XX.X (XX.X) | .X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X(XX.X) |
| Above Normal -> Normal | .X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X(XX.X) |
| Above Normal -> Above Normal XX.X (XX.X) | .X (XX.X) | XX.X(XX.X) | XX.X (XX.X) | XX.X (XX.X) |

Day 2

Etc.

<Programming Note: Continue for Days 3, 4, 6, 10, 14, 17, 20, and 26. Use "—" to indicate not applicable for specific cohorts.>

Note: Baseline is the last available measurement prior to the first dose of the study drug on Day 1.

Generated on XX/XX/XX:XXXX by XXX / Uses: XXXX / Reference: Data Listing XXXX

[Programming Note: For hematology differential, please include only absolute values (not the % for differentials).]


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002

Page X of Y

Table 14.3.2.3.X: Summary of Laboratory Values Outside of Normal Range and Investigator's Assessment [Hematology][ Chemistry][Coagulation] Safety Population

| | TBI-223<br>1800 mg<br>(N=XX) | TBI-223<br>2400 mg<br>(N=XX) | TBI-223<br>3000 mg<br>(N=XX) | Pooled<br>Placebo<br>(N=XX) |
|---|---|---|---|---|
| Number of Subjects with Findings, N (%) | | | | |
| Not clinically significant | XX.X (XX.X) | XX.X(XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Clinically significant | XX.X (XX.X) | XX.X(XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| [Lab Tests Name (Units)] | | | | |
| Number of Subjects with Abnormality, N (%) | XX.X(XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Below Normal | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Above Normal | XX.X(XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X(XX.X) |

Note: Baseline is the last available measurement prior to the first dose of the study drug on Day 1. This summary includes results from any post-baseline visit.

Page X of Y

Table 14.3.2.4.1: Summary of 12-Lead ECG Numeric Results Absolute Values and Change from Baseline by Treatment and Time Point Safety Population

| | TBI-223<br>1800 mg<br>(N=XX) | TBI-223<br>2400 mg<br>(N=XX) | TBI-223<br>3000 mg<br>(N=XX) | Pooled Placebo (N=XX) |
|---|---|---|---|---|
| [Tests Name (Units)] Baseline | | | | |
| Z | × | X | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX | XX |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX | XX, XX |
| Day 1 Post-Dose [2] | | | | |
| Z | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX | XX |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX | XX, XX |
| Change from Baseline | | | | |
| Z | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | X | XX | XX | XX |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX | XX, XX |

<Continue for Days 4, 5-10, 12-17, 18-19, 20, 26>

Note: Baseline is the last available measurement prior to the first dose of the study drug on Day 1.

Generated on XX/XX/XX:XXXX by XXX / Uses: XXXX / Reference: Data Listing XXXX

[Programming note: Summarize all ECG tests with continuous results, including ventricular rate, PR, QRS, QT, QTcF intervals. Page break between ECG tests.]

Page X of Y

Table 14.3.2.4.2: Summary of 12-Lead ECG Categorical Analysis

Safety Population

| | TBI-223<br>1800 mg<br>(N=XX) | TB1-223<br>2400 mg<br>(N=XX) | TBI-223<br>3000 mg<br>(N=XX) | Pooled<br>Placebo<br>(N=XX) |
|---|---|---|---|---|
| QTcF (msec) | | | | |
| Absolute Values [1] | | | | |
| > 450 | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| > 480 | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| > 500 | XX(XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| Change from baseline [2] | | | | |
| > 30 | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| 09 < | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Baseline is the last available measurement prior to the first dose of the study drug on Day 1.

[1] Subjects with QTcF absolute values > (450, 480 and 500 msec) at any post dosing time point are included. [2] Subjects with QTcF change from baseline values > (30 and 60 msec) at any post dosing time point are included. <a href="#"></a>-Programming Note: Additional QTcF value categories may be added to aid data interpretation.


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002

Table 14.3.2.5: Summary of Vital Signs Absolute Values and Change from Baseline by Treatment and Time Point Safety Population

| | TBI-223<br>1800 mg<br>(N=XX) | TBI-223<br>2400 mg<br>(N=XX) | TBI-223<br>3000 mg<br>(N=XX) | Pooled<br>Placebo<br>(N=XX) |
|---|---|---|---|---|
| [Vital Sign Tests Name (Units)] Baseline [1] | X | X | X | X |
| Mean (SD)<br>Median | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX | XX, XX |
| Day 1, 1 Hour Post-Dose | | | | |
| Z | XX | XX | XX | XX |
| Mean (SD)<br>Median | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX | XX, XX |
| Change from Baseline<br>N | * | \$ | XX | * |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX | XX |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX | XX, XX |

<Day 2>

<Day 3>

Note: Baseline is the last available measurement prior to the first dose of the study drug on Day 1.

Page X of Y

Table 14.3.2.5: Summary of Vital Signs
Absolute Values and Change from Baseline by Treatment and Time Point
Safety Population

| ose> | XX XX XX | XX.X(XX.X) $XX.X(XX.X)$ | XX | ımum XX, XX XX, XX XX, XX XX, XX | 90 | XX | XX.X (XX.X) | XX | XX, XX XX, XX | 1 Pre-Dose | XX | XX.X (XX.X) | XX | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <day 14="" 17="" day="" pre-dose=""> Day 14 6 Hours Post-Dose</day> | Z | Mean (SD) | Median | Minimum, Maximum | Change from Baseline | Z | Mean (SD) | Median | Minimum, Maximum | Change from Day 14 Pre-Dose | Z | Mean (SD) | Median | Minimum, Maximum | ; | <day 15=""></day> | <day 16=""></day> |

Note: Baseline is the last available measurement prior to the first dose of the study drug on Day 1.

<Follow-up Visits>


## Sample Figure (same layout for all figures)

Global Alliance for TB Drug Development

Protocol Number: TBI-223-CL-002

Figure 14.2.A.1.1.1: Mean TBI-223 Plasma Concentration by Treatment and Time Point, Linear Scale Hours 0 to 24 Post-Dose, Days 1 (fasted), 4 (fed), and 17 (steady state) Cohort 1, PK Population



Generated on <date-time> by <Program Name> / Uses: <List datasets>

Sample SAS Code (same layout for all figures)

DATA BLANK;

BLANK="";

## Global Alliance for TB Drug Development Protocol No. TBI-223-CL-002 TKL No. P1980121

```
LEGEND1 DOWN=3 POSITION=(TOP RIGHT INSIDE) VALUE=(HEIGHT=2 "Day 1 (fasted)" "Day 4 (fed)" "Day 17 (steady state)") MODE=PROTECT
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                  AXISI LABEL= (ANGLE=90 HEIGHT=2 "Plasma Concentration (mg/L)") ORDER=(0 TO 15 BY 1) VALUE=(HEIGHT=2) MINOR=NONE;
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                      LINE "\par\qc{Figure 14.2.1: Mean TBI-223 Plasma Concentration by Treatment and Time Point, Linear Scale}";
                                                                              ODS RTF FILE="[FILENAME.RTF]" STYLE=STYLES.TEST headery=720 footery=720 nogtitle nogfootnote bodytitle;
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                        COMPUTE AFTER /style=[protectspecialchars=off];
LINE "\q1{ }\brdrt\brdrt\brdrs{}Generated on <date-time> by <Program Name> / Uses: <List datasets>";
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                      AXIS2 LABEL=(HEIGHT=2 "Time Post-dose (h)") VALUE=(HEIGHT=2) ORDER=(0 TO 24 by 2) MINOR=NONE;
                                                                                                                                                                                                                                                                                                                                                                                                                                                               OMPUTE BEFORE PAGE /style=[protectspecialchars=off];
LINE "\q1\b{Global Alliance for TB Drug Development}\b0\tqr\tx12250\tab{}";
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                        GOPTIONS RESET=ALL DEVICE=EMF FTEXT="Albany AMT" HSIZE=6 VSIZE=3.75;
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                       PLOT Y*X=DAY / VAXIS=AXIS1 HAXIS=AXIS2 LEGEND=LEGEND1;
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                             LINE=1 INTERPOL=JOIN;
LINE=5 INTERPOL=JOIN;
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                   SYMBOL1 VALUE=DIAMOND COLOR="BLACK" LINE=20 INTERPOL=JOIN;
                                                                                                                                                                                                                             PROC REPORT DATA=BLANK NOWD SPLIT=" | " MISSING NOCENTER
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                      PROC REPORT DATA=BLANK NOWD SPLIT="|" MISSING NOCENTER
                                                                                                                                                                                                                                                                                                                           STYLE (COLUMN HEADER) = [PROTECTSPECIALCHARS=OFF];
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                STYLE (COLUMN HEADER) = [PROTECTSPECIALCHARS=OFF];
OPTION LS=200 NODATE NONUMBER MISSING=' ';
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                             LINE "Protocol Number: TBI-223-CL-002";
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                   line "Cohort 1, PK Population";
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                            LINE "\par\q1{ }\brdrb\brdrs";
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                              / DISPLAY " ;
                                                                                                                                                                                                                                                                                                                                                                                                                     / DISPLAY " ;
                                                                                                                                                                                                                                                                       STYLE (REPORT) = {OUTPUTWIDTH=8.75in}
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                   STYLE (REPORT) = {OUTPUTWIDTH=8.75in}
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                SYMBOL2 VALUE=CIRCLE COLOR="BLUE"
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                      SYMBOL3 VALUE=SQUARE COLOR="RED"
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                           FORMAT DAY D.;
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                        PROC GPLOT DATA=PLOT;
                                                                                                                                       ODS LISTING CLOSE;
                                                                                                                                                                                                                                                                                                                                                                            COLUMNS BLANK;
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                     COLUMNS BLANK;
                                                                                                                                                                                                                                                                                                                                                                                                                                                                      COMPUTE BEFORE
                                                                                                                                                                                                                                                                                                                                                                                                                     DEFINE BLANK
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                              DEFINE BLANK
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                        LABEL=NONE;
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                     ENDCOMP;
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                      ENDCOMP;
```

Page X of Y

16.1.7: Subject Enrollment and Randomization

All Subjects

| ubject | Subject Date of Informed Consent | Satisfy All I/E<br>Criteria? | Date of<br>Randomization | Randomization<br>Number | Planned<br>Treatment | Actual<br>Treatment |
|---|---|---|---|---|---|---|
| XXX | XX-XX-XXXX | XX | XX-XX-XXXX | XXXXXX | XXXX | XXXX |
| XXX | XX-XX-XXX | XX | XX-XX-XXXX | XXXXX | XXXX | XXXX |
| 001 | 2020-06-19 | Yes | 2020-07-08 | 0345 | TBI-223 1800mg | TBI-223 1800mg |

Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002

| | 1201 | 2717 |
|-------|-------|------|
| : | - | Ę |
| r | Ç | 3 |
| | 70002 | 2 |
| | 3 | 2 |
| ζ | / | 2 |
| _ | • | : |
| ٦ | | • |
| ٦ | | : |
| ( | | i |
| 0 / - | ٥ | 2 |
| 7 | | _ |

| Date of<br>Subject Informed<br>Consent | Date of<br>Screening | Ethnicity | Gender Race | Serious Adverse Event<br>Reported? | Inclusion/Exclusion<br>Criteria Not Met | Additional Reason for<br>Screen Failure |
|---|---|---|---|---|---|---|
| | -XX-XXX | | | | | |
| XX-XX-XXXX XXX | XX | XXX | XXX XXX | XXX | XXXX | XXXX |
| | XXXXX-XX | | | | | |
| XX-XX-XXXX XXX | XX | XXX | XXX XXX | XXX | XXXX | XXXX |
| 5002 2020-06-19 | 2020-06-19 | 2020-06-19 Hispanic or Latino Female White | no Female White | No | Inclusion 3 | : |

Generated on XX/XX/XX:XXXXXXXX by XXXX/ Uses: XXXX

[Programming Note: Include all additional reasons for screen failure and display format "Other: XXXXXX". XXXX is the detailed reason. Use semi-colon to separate each reason.]


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002

16.2.1.2: Disposition of Subjects

All Randomized Subjects

[TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

| | | | Date (Day) of [1] | y) of [1] | | | |
|---|---|---|---|---|---|---|---|
| Subject | Screening | Randomization | First Dose | Last Dose | Last Visit | Last Contact | Study Completion<br>Status |
| XXX | XXXXX-XXX- | -XX-XXX | -XX-XXX | XXXXX-XXX- | XXXX-XXX- | XXXX-XXX- | XXXXX |
| | XX(XX) | XX(XX) | XX(XX)<br>TXX:XX | XX(XX)<br>TXX:XX | XX(XX) | XX(XX) | |
| XXX | XXXX-XX-<br>XX(XX) | XXXXX-XX-<br>XX(XX) | XXXX-XX-XX-XX-XX-XX-XX-XX-XX-XX-XX-XX-X | XXXXX-XX-XX-XXX-XXX | XXXX-XX-<br>XX(XX) | XXXX-XX-XX-XX-XXX | XXXXX |
| 0120 | 2020-06-19 (-10) | 2020-06-29 (1) | TXX:XX<br>2020-06-29 (1)<br>T08:30 | XXXXX-XX-<br>XX(XX)<br>XX(XX)<br>TXX:XX | 2020-07-06(8) | XXXXX-XX-XX-XX-XX-XX-XX-XX-XX-XX-XX-XX- | Completed |

[1] Day is calculated relative to Day 1.

Generated on XX/XX/XX:XXXX by XXXX/ Uses: XXXX

[Programming Note: Study completion status will include reason for discontinuation if a subject does not complete the study.]

Global Alliance for TB Drug Development Protocol No. TBI-223-CL-002 TKL No. P1980121 Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002 16.2.2: Protocol Deviation Safety Population [TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

| | Action Taken | XXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|---|---|---|
| | Protocol Deviation Type | XXXXXXXX | XXXXXXXX |
| | Protocol Deviation | XXXX | XXXX |
| | Visit (Date) | XX (XX-XX-XXX) | XX (XX-XX-XXXXX) |
| Major or | Subject Minor | Major | Minor |
| | Subject | XXX | |

Generated on XX/XX/XX:XXXX by XXXX/ Uses: XXXX

[Programming Note: If site deviation or deviation for SF subjects are also available, include those at the very end of this listing.]


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002 16.2.3: Population Datasets

[TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

| Subject | In Safety Population? | In PK Population? |
|---------|-----------------------|-------------------|
| XXX | Yes<br>No | Yes<br>No |


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002

16.2.4.1: Demographics and Baseline Characteristics [TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

Safety Population

| BMI (kg/m²) [1] | XXX.X | XX.X |
|-----------------|-----------------|-----------------|
| Height (cm) | XXX | XXX |
| Weight (kg) | XXX | XXX |
| Ethnicity | XX | XX |
| Race | XXXX | XXXX |
| Gender | Male | Female |
| Age (years) Ger | XX | XX |
| Cohort | TBI-223 1800 mg | TBI-223 1800 mg |
| Subject | XXX | XXX |

Note: BMI = Body Mass Index [1] Baseline BMI is calculated as baseline weight / baseline height^2.

Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002 16.2.4.2: Prior and Concomitant Medication

[TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

Safety Population

| Subject | Prior or<br>Concomitant? | WHO Preferred Term (Verbatim Term) Prior or / Subject Concomitant? ATC Classification | Indication<br>Dose Unit/Frequency/Route | Start Date (Day)-Stop Date (Day) |
|---|---|---|---|---|
| XXX | Concomitant | Concomitant XXXXXX (xxxxx)/ XXXXXXX | XXX<br>XX XX/XXX/XXXX | XXXX-XXX (XX) – XXXX-XX-XXX-XXX-XXX (XX) |
| XXX | Concomitant | XXXXXX/<br>XXXXXXX | XXX<br>XX XX/XXX/XXXX | DNIODNO – (XX) XX-XX-XXXX |

Generated on XX/XX/XX:XXXX by XXXX/ Uses: XXXX

[Programming Note: List medication in ascending start date for each subject.]


Page X of Y

16.2.4.3: Medical and Surgical History

[[TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

Safety Population

| Subject | Diagnosis / Procedure | Start Date (Day) | End Date (Day) | Medication Taken Currently? |
|---|---|---|---|---|
| XXXX | XXXX | (XX) XX-XX-XXXX | XXXXX-XXX (XX) | no |
| | XXXX | XXX-XX-XXX (XX) | ONGOING | yes |


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002 16.2.5.1: Plasma Concentrations [TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg] Safety Population

| g/mL) | M2 | XX.X | XX.X | XXX.X | XX.X |
|---|---|---|---|---|---|
| Concentration (ng/mL) | TBI-223 | XX.X | XX.X | XX.X | XX.X |
| - | Elapsed<br>Time (h) | XX,X | XX,X | XX,X | XX,X |
| | Sample Collection<br>Date and Time (Day) | XXXX-XX-XX TXX:XX (XX) | XXXXX-XX-XX TXX:XX (XX) | XXXXX-XX-XX TXX:XX (XX) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | Date and Time (Day) | XXXXX-XX-XX TXX:XX (XX) | | | |
| | Subject Visit PK Time Point | Pre-dose | 30 min | 1 hour | <etc.></etc.> |
| | Visit | Day 1 | | | <etc.></etc.> |
| | Subject | XXX Day 1 | | | |


| Protocol Nu | Otobal Alliance for 1.B Drug Devel<br>Protocol Number: TBI-223-CL-002 | Global Alliance for 1 B Drug Development<br>Protocol Number: TBI-223-CL-002 | nt | | | | | | | | rage A 01 1 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | П | 16.2.5.2: 7<br>[TBI-2 | ГВІ-223<br>223 1800 | Pharmac<br>)mg][TB | 5.2: TBI-223 Pharmacokinetic Param<br>[TBI-223 1800mg][TBI-223 2400mg] | 16.2.5.2: TBI-223 Pharmacokinetic Parameters [TBI-223 1800mg][TBI-223 2400mg] | | | |
| | | | | | PK | PK Population | ion | | | | |
| Subject | Visit | $	ext{AUC}_{0.24}$ (µg.h/mL) | AUCinf<br>(μg.h/mL) | C <sub>max</sub> (µg) | T <sub>max</sub><br>(h) | Cmin<br>(µg) | $\Gamma_{min}$ $(h)$ | CL/F (L/h) | $V_{z}/F(L)$ | RAUC | RCmax |
| XXX | Day 1 | XXX | XXX | XXX | XXX | 1 | ; | XXX | XXXX | 1 | 1 |
| | Day 4 | XXX | XXX | XXX | XXX | ł | ł | XXX | XX.XX | 1 | 1 |
| | Day 17 | XXX | ł | XXX | XXX | XXX | XXX | 1 | ŀ | X.XXX | X.XXX |
| Generated on | XX/XX/XX | Generated on XX/XX/XX:XXXX by XXXX/ Uses: XXXX | 7 Uses: XXXX | | | | | | | | |
| Global Allia<br>Protocol Nu | Global Alliance for TB Drug Devel<br>Protocol Number: TBI-223-CL-002 | Global Alliance for TB Drug Development<br>Protocol Number: TBI-223-CL-002 | nt | | | | | | | | Page X of Y |
| | | | 1 | 16.2.5.2: 7 | rbi-223<br>Tbi | 223 Pharmacokine<br>TBI-223 3000mg | okinetic l<br>0mg | 16.2.5.2: TBI-223 Pharmacokinetic Parameters<br>TBI-223 3000mg | | | |
| | | | | | PK | PK Population | ion | | | | |
| Subject | Visit | AUC <sub>0-24</sub><br>(μg.h/mL) | AUCinf<br>(μg.h/mL) | С <sub>max</sub><br>(µg) | T <sub>max</sub> (h) | Cmin<br>(µg) | $T_{min}$ (h) | CL/F (L/h) | $ m V_z/F$ (L) | RAUC | RCmax |
| XXX | Day 1 | XXX | XXX | XXX | XXX | 1 | 1 | XXX | XX.XX | ŀ | ł |
| | Day 14 | XXX | 1 | XXX | XXX | XXX | XXX | 1 | 1 | X.XXX | X.XXX |


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002 16.2.5.3: TBI-223 Elimination Rate Constant and Half-Life [TBI-223 1800mg][TBI-223 2400mg]

| | | | J | | | | |
|---|---|---|---|---|---|---|---|
| Subject | Visit | Start Time of Elimination<br>Phase (h) | limination End Time of Elimination<br>h) Phase (h) | Number of Points<br>Included | $\lambda z (h^{-1})$ | t <sub>1/2</sub> (h) | $\lambda z (h^{-1})$ $t_{1/2} (h)$ R-square |
| | | - | | 1 | c | | |
| YYY | Day 1 | XX | XX | × | U.XXX | X.XX | U.XXX |
| | Day 4 | XX | XX | × | 0.xxx | X.XX | 0.xxx |
| | Day 17 | XX | XX | × | 0.xxx | X.XX | 0.xxx |
| XXX | Day 1 | XX | XX | × | 0.xxx | X.XX | 0.xxx |
| | Day 4 | XX | XX | × | 0.xxx | X.XX | 0.xxx |
| | Day 17 | XX | XX | × | 0.xxx | x.xx | 0.xxx |


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002 16.2.5.3: TBI-223 Elimination Rate Constant and Half-Life TBI-223 3000mg

| | R-square | 0.xxx<br>0.xxx | 0.xxx<br>0.xxx |
|---|---|---|---|
| | $\lambda z (h^{-1})$ $t_{1/2} (h)$ R-square | X.XX<br>X.XX | X.XX<br>X.XX |
| | λz (h <sup>-1</sup> ) | 0.xxx<br>0.xxx | 0.xxx<br>0.xxx |
| | Number of Points<br>Included | ×× | × × |
| PK Population | limination End Time of Elimination<br>h) Phase (h) | X X | XX XX |
| | Start Time of Elimination<br>Phase (h) | XX XX | XX |
| | Visit | Day 1<br>Day 14 | Day 1<br>Day 14 |
| | Subject | XXX | XXX |


| Global Alli:<br>Protocol Nu | Global Alliance for TB Drug Devel<br>Protocol Number: TBI-223-CL-002 | Global Alliance for TB Drug Development<br>Protocol Number: TBI-223-CL-002 | ıt | | | | | | | | Page X of Y |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 16.2.5.4<br>[TBI-3 | : M2 Phz<br>223 1800 | armacoki<br>mg][TB | 16.2.5.4: M2 Pharmacokinetic Parameters [TBI-223 1800mg][TBI-223 2400mg] | ameters<br>)0mg] | | | |
| | | | | | PK | PK Population | ion | | | | |
| Subject | Visit | AUC <sub>0-24</sub><br>(μg.h/mL) | AUC <sub>inf</sub><br>(μg.h/mL) | Стах (µg) | T <sub>max</sub> (h) | Cmin (µg) | T <sub>min</sub> (h) | CL/F (L/h) | $V_z/F(L)$ | RAUC | RCmax |
| XXX | Day 1 | XXX | XXX | XXX | XXX | 1 | 1 | XXX | XX.XX | ŀ | ł |
| | Day 4 | XXX | XXX | XXX | XXX | 1 | ł | XXX | XX.XX | 1 | ŀ |
| | Day 17 | XXX | ŀ | XXX | XXX | XXX | XXX | 1 | ŀ | X.XXX | X.XXX |
| Generated or | XX/XX/XX: | Generated on XX/XX/XX:XXXX by XXXX/ Uses: XXXX | / Uses: XXXX | | | | | | | | |
| Global Alli:<br>Protocol Nu | Global Alliance for TB Drug Devel-<br>Protocol Number: TBI-223-CL-002 | Global Alliance for TB Drug Development<br>Protocol Number: TBI-223-CL-002 | ıt | | | | | | | | Page X of Y |
| | | | | 16.2.5.4 | : M2 Pha<br>TBI | Pharmacokinetic<br>TBI-223 3000mg | 16.2.5.4: M2 Pharmacokinetic Parameters<br>TBI-223 3000mg | ameters | | | |
| | | | | | PK | PK Population | ion | | | | |
| Subject | Visit | AUC <sub>0-24</sub><br>(μg.h/mL) | AUCinf<br>(μg.h/mL) | Стах (µg) | T <sub>max</sub> (h) | Cmin (µg) | T <sub>min</sub> (h) | CL/F (L/h) | $V_z/F(L)$ | RAUC | RCmax |
| XXX | Day 1 | XXX | XXX | XXX | XXX | 1 | ŀ | XXX | XX.XX | ; | ł |
| | Day 14 | XXX | 1 | XXX | XXX | XXX | XXX | ŀ | ŀ | X.XXX | X.XXX |


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002 16.2.5.5: M2 Elimination Rate Constant and Half-Life [TBI-223 1800mg][TBI-223 2400mg]

| | t <sub>1/2</sub> (h) R-square | 0.xxx | 0.xxx | 0.xxx | 0.xxx | 0.xxx | 0.xxx |
|---|---|---|---|---|---|---|---|
| | | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | $\lambda z (h^{-1})$ | 0.xxx | 0.xxx | 0.xxx | 0.xxx | 0.xxx | 0.xxx |
| | Number of Points<br>Included | × | X | × | × | X | × |
| PK Population | Elimination End Time of Elimination (h) | XX | XX | XX | XX | XX | XX |
| | Start Time of Elimination<br>Phase (h) | XX | XX | XX | XX | XX | XX |
| | Visit | Day 1 | Day 4 | Day 17 | Day 1 | Day 4 | Day 17 |
| | Subject | XXX | | | XXX | | |


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002

16.2.5.5: M2 Elimination Rate Constant and Half-Life TBI-223 3000mg

| | R-square | 0.xxx | 0.xxx | 0.xxx<br>0.xxx |
|---|---|---|---|---|
| | λz (h-1) t <sub>1/2</sub> (h) R-square | X.XX | X.XX | X.XX<br>X.XX |
| | $\lambda z \left( h^{-1} \right)$ | 0.xxx | 0.xxx | 0.xxx<br>0.xxx |
| | Number of Points<br>Included | × | × | × × |
| PK Population | Elimination End Time of Elimination (h) Phase (h) | XX | XX | x x |
| | Start Time of Elimination<br>Phase (h) | XX | XX | X X |
| | Visit | Day 1 | Day 14 | Day 1<br>Day 14 |
| | Subject | XXX | | XXX |


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002

16.2.5.6: Fasting and Meals [TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

PK Population

| Fast 4 hour duration post-<br>dosing | Yes<br>Yes |
|---|---|
| Breakfast end within 5 min Fast 4 prior to dosing | Yes<br>Yes |
| | Yes<br>Yes |
| Fast 10 hours duration prior to Standard Breakfast 30 min dosing | Yes<br>Yes |
| | Day 1<br>Etc. |
| Subject Visit | XXX |

Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002

16.2.7.1: Adverse Events [TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

Safety Population

| Subject | MedDRA Preferred Term<br>(Verbatim Term) /<br>Subject MedDRA SOC Term | Start Date (Day)and Time -<br>End Date (Day) and Time | TEAE? [1] / Severity/ Outcome/ Relationship [2] | Action Taken with Study Product<br>Other Action Taken /<br>Serious (Which Criteria Met)? |
|---|---|---|---|---|
| XXX | XXXXXXX | - XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Yes/ | Not Applicable/ |
| | (XXXXXX)/ | XXXXX-XXX-XXX | Mild/ | Concomitant Medication / |
| | XXXXXXXXX | | Recovered/Resolved/ | Yes (Hospitalization) |
| | | | Not Related | |
| | XXXXXXX | - XXX:XXX (XX) XXX-XXX | Yes/ | Not Applicable / |
| | (XXXXXX)/ | XXXXX-XXX-XXX | Mild/ | None / |
| | XXXXXXXXX | | Recovered/Resolved/ | No |
| | | | Possible | |

[1] TEAE is defined as an AE with a start date and time on or after the first dose of any study drugs. [2] Relationship is determined by the Investigator between an AE and the study drug unless otherwise specified.

Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002 16.2.7.2: Serious Adverse Events and Adverse Events Leading to Study Discontinuation [TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

## Safety Population

| Subject | MedDRA Preferred Term<br>(Verbatim Term) /<br>Subject MedDRA SOC Term | Start Date (Day)and Time -<br>End Date (Day) and Time | TEAE? [1] / Severity/ Outcome/ Relationship [2] | Action Taken with Study Product<br>Other Action Taken /<br>Serious (Which Criteria Met)? |
|---|---|---|---|---|
| XXX | XXXXXXX<br>(XXXXXXX)/<br>XXXXXXXXXX | XXXXX-XX-XX (XX) TXX:XX – XXXX-XXX (XX) TXX:XX | Yes/<br>Mild/<br>Recovered/Resolved/<br>Not Related | Drug Reduced /<br>Concomitant Medication /<br>Yes (Hospitalization) |
| | XXXXXXX<br>(XXXXXX)/<br>XXXXXXXXXX | XXXX-XX-XX (XX) TXX:XX – XXXX-XX (XX) TXX:XX | Yes/<br>Mild/<br>Recovered/Resolved/<br>Probable | Drug Withdrawn / Discontinued Study / Yes (Life Threatening) |

<sup>[1]</sup> TEAE is defined as an AE with a start date and time on or after the first dose of any study drugs. [2] Relationship is determined by the Investigator between an AE and the study drug unless otherwise specified.

Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002

Page X of Y

16.2.8.1: Childbearing Potential and Serum Pregnancy Tests [TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

Safety Population

| Result | Negative<br>Negative |
|------------------------|-------------------------------------|
| Date (Day) | (XX) XX-XX-XXXX<br>XXXX-XX-XXX (XX) |
| Visit | Screening<br>Day -2 (Check-In) |
| Childbearing Potential | IUD |
| Subject | XXX |


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002

16.2.8.2: Urine Drug and Alcohol Screenings [TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

Safety Population

| Subject | Visit | Date (Day) | Urine Drug Screen | Urine Alcohol Screen | Urine Cotinine Screen |
|---|---|---|---|---|---|
| XXX | Screening | XXXX-XX-XX(XX) | Negative | Negative | Negative |
| | Day -2 (Check-In) | XXXX-XX-XX (XX) | Negative | Negative | Negative |


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002 16.2.8.3: Clinical Laboratory Tests – Investigator's Assessments [TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

Investigator's Assessment Abnormal NCS Normal Normal Normal Serum chemistry Lab Category Hematology Coagulation Urinalysis Safety Population Date and Time (Day) Etc. Screening Day -1 Visit Subject XXX

Note: NCS = Not clinically significant. CS = Clinically significant.

Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002 [Serum Chemistry][Hematology][Urinalysis][Coagulation] [TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

Safety Population

| Subject | Subject Visit | Date and Time (Day) | Parameter<br>(Unit) | Reference Range | Result /<br>Abnormality | CFBL[1] |
|---|---|---|---|---|---|---|
| XXX | Screening Day -1 Day 1 Etc. | XXXX-XX-XXTXX:XX (XX)<br>XXXX-XX-XXTXX:XX (XX)<br>XXXX-XX-XXTXX:XX (XX) | XXXX | XXXX,XXXX | XXXX<br>XXXX/L<br>XXXX/H | XXXXX<br>XXXXX<br>XXXXX |

Note: H = High; L = Low. A = Abnormal, unspecified high or low.

[1] CFBL = Change from Baseline. Baseline value is the last available measurement prior to first dose of study drug.

Generated on XX/XX/XX:XXXX by XXXXX / Uses: XX

[Programming Note: Urinalysis will not have CFBL column. Include all available visits. For out of range results, add a letter (A, H or L) in bold right next the results.]


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002

16.2.8.5: Laboratory Values Outside of Normal Range [TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

Safety Population

| Reference Range XXXX,XXXX XXXX,XXXX | | | | | Parameter | | | |
|---|---|---|---|---|---|---|---|---|
| Day -1XXXX-XX-XX-XXTXX:XX (XX)ChemistryXXXXXXXXX,XXXXDay -1XXXX-XX-XX-XXTXX:XX (XX)HematologyXXXXXXXXX | Subject | Visit | | Category | (Unit) | Reference Range | Result | Abnormality |
| | XXX | | XXXXX-XX-XXTXX:XX (XX)<br>XXXX-XX-XXTXX:XX (XX) | Chemistry<br>Hematology | XXXX | XXXX,XXXX<br>XXXX,XXXX | XX.XX<br>XX.XX | Low<br>High |


Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002 16.2.8.6: Vital Signs

[TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

Safety Population

| CFBL [1] | I | ; | Baseline | XXX | |
|---|---|---|---|---|---|
| Result | XXX | XXX | XXX | XXX | |
| Parameter (Unit) | Systolic BP (mmHg) | Systolic BP (mmHg) | Systolic BP (mmHg) | Systolic BP (mmHg) | |
| Date and Time (Day) | XXXX-XX-XXTXX:XX (XX) | XXXX-XX-XX-XXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXX-XX-XXTXX:XX (XX) | XXXXX-XX-XXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| Time Point | I | 1 | Pre-dose | 1 Hour Post-dose | |
| Subject Visit | Screening | Day -2 | Day 1 | Day 1 | Etc. |
| Subject | XXX | | | | |

Also include tests: Diastolic BP (mmHg), Pulse Rate (beats/min), Respiration Rate (breaths/min), Temperature (°C), Pulse Oximetry

BP = Systolic Blood Pressure

[1] CFBL = Change from Baseline. Baseline value is the last available measurement prior to first dose of study drug.

Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002 16.2.8.7.1: Physical Examinations [TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

Comment XXXXX All Other Body Systems Normal All Body Systems Normal Abnormal Result Safety Population **Body System** All Other XXX All XXX-XX-XXX Date of Test (Day) (XX) XX-XX-XXX (XX) XX-XX-XXX Screening Day -1 Day -1 Visit Etc. Subject XXX

Note: Body systems examined include Cardiovascular, Respiratory, Gastrointestinal, Musculoskeletal, Skin, Systemic, and Other.

Global Alliance for TB Drug Development

Protocol Number: TBI-223-CL-002

16.2.8.7.2: Neurological Examinations [TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

Safety Population

| Subject | Visit | Date of Test (Day) | Nervous System | Findings | Comment |
|---|---|---|---|---|---|
| XXX | Screening Day -1 Day -1 | (XX) XX-XX-XXX<br>XXX-XX-XX-XXX<br>(XX) XX-XX-XXX | All XXX All Other | All Nervous Systems Normal Abnormal All Other Nervous Systems Normal | - XXXXXX |

Note: Neurological systems examined include Mental Status: Orientation, Speech, and Memory, Cranial Nerves 2 through 12, Motor System, Sensory System: Face, Neck, Arms, Trunk, and Legs, Reflexes. Coordination: Upper Body and Lower Body, Gait, and Other.

Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002 16.2.8.8: 12-Lead ECG Results [TBI-223 1800mg][TBI-223 3000mg][Pooled Placebo]

Safety Population

| Subject | Visit | Date and Time (Day) | Investigator's Assessment | Test (Unit) Result CFBL [1] | Result | CFBL [1] |
|---|---|---|---|---|---|---|
| XXX | Screening | XXXXX-XXX-XXXXXXXXXXXXXXXXXXXXXXXXXXXX | Normal | Heart Rate | XXX | XXX |
| | | | | PR Interval | XXX | XXX |
| | | | | Etc. | XXX | XXX |
| | Day 1 Pre-dose | XXXX-XX-XXTXX:XX (XX) | Normal | Heart Rate | XXX | XXX |
| | | | | PR Interval | XXX | XXX |
| | | | | Etc. | XXX | XXX |
| | Etc. | | | | | |

[1] CFBL = Change from Baseline. Baseline value is the last available measurement prior to first dose of study drug.

Generated on XX/XX/XX:XXXX by XXXX / Uses: XXXX

[Programming Note: Include all visits and all ECG tests collected on the CRF (ventricular rate, PR, QRS, QT, QTcF).]

Global Alliance for TB Drug Development Protocol No. TBI-223-CL-002 TKL No. P1980121 Global Alliance for TB Drug Development Protocol Number: TBI-223-CL-002 16.2.9: General Comments

[TBI-223 1800mg][TBI-223 2400mg][TBI-223 3000mg][Pooled Placebo]

Safety Population

| Comment | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|-------------------|-----------------------------------------|
| Comment Reference | XXXX<br>XXXX |
| Subject | XXX |



# **Certificate Of Completion**

Envelope Id: B5BB91B52BEB41D0993F26E00A6EAA0E

Subject: Please DocuSign: tbi-223-cl-002-mad-sap-final-2021-03-24 - unsigned.pdf

Source Envelope:

Document Pages: 82 Signatures: 2 **Envelope Originator:** Certificate Pages: 5 Initials: 0 Marie Messina AutoNav: Enabled 40 Wall St FL 24 Envelopeld Stamping: Disabled New York, NY 10005

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

marie.messina@tballiance.org IP Address: 184.152.37.209

Sent: 20 April 2021 | 10:58

Viewed: 20 April 2021 | 11:07

Signed: 20 April 2021 | 11:07

Status: Completed

#### **Record Tracking**

Status: Original Holder: Marie Messina Location: DocuSign

20 April 2021 | 10:55 marie.messina@tballiance.org

| Signer Events | Signature | Timestamp |
|---|---|---|
| Jerry Nedelman | | Sent: 20 April 2021 10:58 |
| jerry.nedelman@tballiance.org | Jerry Medelman | Viewed: 20 April 2021 11:04 |
| Senior Director, Pharmacometrics | | Signed: 20 April 2021 11:04 |
| Security Level: Email, Account Authentication (Required) | Signature Adoption: Pre-selected Style Signature ID: 7839E5A7-6523-498A-B928-E27ED5F738EA Using IP Address: 71.187.221.226 | |
| | With Signing Authentication via DocuSign passwo | ord |
| | With Signing Reasons (on each tab): | |

I have reviewed this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 06 September 2017 | 09:47 ID: 14a4057c-d83c-405f-bceb-b7e7952cc709

Michael Tuley

mtuley@tklresearch.com

Michael TKL

Security Level: Email, Account Authentication

(Required)

Michael Tuley

Signature Adoption: Pre-selected Style

Signature ID:

BE981D7A-3194-4349-9E30-D520D1EBB3FD

Using IP Address: 70.36.31.130

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 20 January 2021 | 15:54 ID: 63f91ddf-4564-4029-968b-d91f4c9fbc68

| In Person Signer Events | Signature | Timestamp |
|------------------------------|-----------|-----------|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |

| Carbon Copy Events | Status | Timestamp |
|---|---|---|
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 20 April 2021 10:58 |
| Certified Delivered | Security Checked | 20 April 2021 11:07 |
| Signing Complete | Security Checked | 20 April 2021 11:07 |
| Completed | Security Checked | 20 April 2021 11:07 |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disc | losure | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Global Alliance for TB Drug Development-Sub Account (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through your DocuSign, Inc. (DocuSign) Express user account. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to these terms and conditions, please confirm your agreement by clicking the 'I agree' button at the bottom of this document.

# **Getting paper copies**

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. For such copies, as long as you are an authorized user of the DocuSign system you will have the ability to download and print any documents we send to you through your DocuSign user account for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

# Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. To indicate to us that you are changing your mind, you must withdraw your consent using the DocuSign 'Withdraw Consent' form on the signing page of your DocuSign account. This will indicate to us that you have withdrawn your consent to receive required notices and disclosures electronically from us and you will no longer be able to use your DocuSign Express user account to receive required notices and consents electronically from us or to sign electronically documents from us.

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through your DocuSign user account all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

### How to contact Global Alliance for TB Drug Development-Sub Account:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: christi.baine@tballiance.org

# To advise Global Alliance for TB Drug Development-Sub Account of your new e-mail address

To let us know of a change in your e-mail address where we should send notices and disclosures electronically to you, you must send an email message to us at christi.baine@tballiance.org and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.. In addition, you must notify DocuSign, Inc to arrange for your new email address to be reflected in your DocuSign account by following the process for changing e-mail in DocuSign.

To request paper copies from Global Alliance for TB Drug Development-Sub Account To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an e-mail to christi.baine@tballiance.org and in the body of such request you must state your e-mail address, full name, US Postal address, and telephone number. We will bill you for any fees at that time, if any.

To withdraw your consent with Global Alliance for TB Drug Development-Sub Account To inform us that you no longer want to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your DocuSign account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send us an e-mail to christi.baine@tballiance.org and in the body of such request you must state your e-mail, full name, IS Postal Address, telephone number, and account number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

Required hardware and software

| Operating Systems: | Windows2000? or WindowsXP? |
|----------------------------|----------------------------------------------|
| Browsers (for SENDERS): | Internet Explorer 6.0? or above |
| Browsers (for SIGNERS): | Internet Explorer 6.0?, Mozilla FireFox 1.0, |
| | NetScape 7.2 (or above) |
| Email: | Access to a valid email account |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | •Allow per session cookies |
| | Allow per session cookies |
| | •Users accessing the internet behind a Proxy |
| | Server must enable HTTP 1.1 settings via |
| | proxy connection |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an email message at the email address we have on file for you at that time providing you with the revised hardware and software requirements, at which time you will

have the right to withdraw your consent.

# Acknowledging your access and consent to receive materials electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please verify that you were able to read this electronic disclosure and that you also were able to print on paper or electronically save this page for your future reference and access or that you were able to e-mail this disclosure and consent to an address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format on the terms and conditions described above, please let us know by clicking the 'I agree' button below.

By checking the 'I Agree' box, I confirm that:

- I can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC RECORD AND SIGNATURE DISCLOSURES document; and
- I can print on paper the disclosure or save or send the disclosure to a place where I can print it, for future reference and access; and
- Until or unless I notify Global Alliance for TB Drug Development-Sub Account as described above, I consent to receive from exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to me by Global Alliance for TB Drug Development-Sub Account during the course of my relationship with you.